| <b>Document Type:</b> | Statistical Analysis Plan |
|---|---|
| Official Title: | Randomized, Double-Masked, Active-Controlled, Phase 3 Study of the Efficacy and Safety of Aflibercept 8 mg in Macular Edema Secondary to Retinal Vein Occlusion |
| NCT Number: | NCT05850520 |
| <b>Document Date:</b> | 21 NOV 2024 |

Version 2.0 Page: 1 of

# Title Page

Protocol Title: Randomized, Double-Masked, Active-Controlled, Phase 3 Study of the Efficacy and Safety of Aflibercept 8 mg in Macular Edema Secondary to Retinal Vein Occlusion

**Protocol Number: 22153** 

Compound Number: BAY 86-5321/aflibercept

Short Title: Efficacy and Safety of High Dose Aflibercept in Macular Edema Secondary to

**Retinal Vein Occlusion** 

**Acronym:** QUASAR

Sponsor Name: Bayer AG

Legal Registered Address: Bayer AG, 51368 Leverkusen, Germany

**Regulatory Agency Identifier Number(s):** 

Investigational New Drug (IND): 12462 (Regeneron Pharmaceuticals, Inc.)

EU-CT number: 2022-502174-16-00

Date: 21 NOV 2024

Version: 2.0

Statistical Analysis Plan template version: 4.0

#### Confidential

The information provided in this document is strictly confidential and is intended solely for the performance of the clinical investigation. Reproduction or disclosure of this document, whether in part or in full, to parties not associated with the clinical investigation or its use for any other purpose without the prior written consent of the sponsor is not permitted.

Throughout this document, symbols indicating proprietary names (®, TM) may not be displayed. Hence, the appearance of product names without these symbols does not imply that these names are not protected.

This Statistical Analysis Plan is produced on a word-processing system and bears no signatures. The approval of the Statistical Analysis Plan is documented in a separate signature document.

# 

# **Table of Contents**

| Title P | Page | 1 |
|---|---|---|
| <b>Table</b> | of Contents | 2 |
| Tables | s of Tables | 3 |
| Tables | s of Figures | 4 |
| | on History | |
| List of | f Abbreviations | 7 |
| 1. | Introduction | 9 |
| 1.1 | Objectives, Endpoints, and Estimands | 10 |
| 1.2 | Study Design | 16 |
| 2. | Statistical Hypotheses | 18 |
| 2.1 | Multiplicity Adjustment | 19 |
| 3. | Analysis Sets | 21 |
| 4. | Statistical Analyses | |
| 4.1 | General Considerations | |
| 4.1.1 | Definition of Dropouts | |
| 4.1.2 | Handling of Missing Data | |
| 4.1.3 | Data Rules | |
| 4.1.4 | Unscheduled Assessments | 25 |
| 4.1.5 | End of Study / Early Discontinuation Visit | 25 |
| 4.1.6 | Definition of Fellow-Eye Treatment | |
| 4.1.7 | Definition of Prohibited Medications | |
| 4.1.8 | Imaging data assessed by the reading center | |
| 4.2 | Primary Endpoint Analysis | |
| 4.2.1 | Definition of Endpoint | |
| 4.2.2 | Main Analytical Approach | |
| 4.2.3 | Sensitivity Analyses | |
| 4.2.4 | Supplementary Analysis | |
| 4.3 | Secondary Endpoints Analysis | |
| 4.3.1 | Key Secondary Endpoint | |
| 4.3.2 | Supportive Secondary Endpoints | 42 |
| 4.4 | Exploratory Endpoints Analysis | |
| 4.4.1<br>4.4.2 | Change from baseline in BCVA measured by the ETDRS letter score at each Participant with vision changes of at least 5, 10, or 15 letters in BCVA from better the baseline in BCVA from better the base | |
| 4.4.2 | at each visit | |
| 4.4.3 | Participant with no IRF and no SRF in the center subfield at each visit | |
| 4.4.4 | Time to fluid-free retina over 36 and 64 weeks (total fluid, IRF, and/or SRF i center subfield) | n the |
| 4.4.5 | Participant having sustained fluid-free retina over 36 and 64 weeks (total fluid and/or SRF in the center subfield) | d, IRF, |
| 4.4.6 | Change in area of retinal ischemia at Weeks 36 and 64 | |
| 4.4.7 | Change in the area of fluorescein leakage at Weeks 36 and 64 | 47 |
| 4.5 | Safety Analyses | 47 |

Version 2.0 

| 4.5.1 | Adverse Events | 47 |
|---|---|---|
| 4.5.2 | Additional Safety Assessments | 49 |
| 4.6 | Other Analyses | |
| 4.6.1 | Subgroup Analyses | 52 |
| 4.6.2 | Subgroup Analysis by RVO type | 53 |
| 4.7 | Interim Analyses and Data Monitoring Committee | |
| 4.8 | Changes to Protocol-planned Analyses | |
| 5. | Sample Size Determination | 54 |
| 6. | Supporting Documentation | 55 |
| 6.1 | Appendix 1: Population characteristics | 55 |
| 6.1.1 | Demographics and baseline characteristics | 55 |
| 6.1.2 | Medical History | 56 |
| 6.1.3 | Exposure and Compliance to Study Intervention | 56 |
| 6.1.4 | Disposition of Study Participants | |
| 6.1.5 | Prior and Concomitant Medication | 59 |
| 6.2 | Appendix 2: Pre-defined Laboratory Abnormalities | 60 |
| 6.3 | Appendix 3: Definition of safety subgroups | 61 |
| 6.3.1 | Hypertension | 61 |
| 6.3.2 | Intraocular inflammation | 62 |
| 6.3.3 | Nasal mucosal events | 62 |
| 6.3.4 | Medical history of cerebrovascular disease (e.g. CVA / Stroke) | 63 |
| 6.3.5 | Medical history of ischaemic heart disease (e.g., myocardial infarction) | 69 |
| 6.3.6 | Medical history of renal impairment | |
| 6.3.7 | Medical history of hepatic impairment | 73 |
| 6.4 | Appendix 4: Handling of Questionnaires | 83 |
| 6.4.1 | NEI-VFQ-25 Sub-scale Scores and Total Score | 83 |
| 6.5 | Appendix 5: Strategies for displaying Summary Statistics | 85 |
| 6.6 | Appendix 6: Identification of intake of prohibited medications and cases of prohibited procedures | |
| | • | |
| 7. | References | 87 |
| Table | es of Tables | |
| Table | 1-1: Objectives and endpoints | 10 |
| | 1-2: Supplementary Estimand for the Primary Objective | |
| | 3-1: Analysis Sets | |
| | 4-1: Number of decimal places for summary statistics | 22 |
| Table 4 | 4-2: Implementation strategies for the handling of intercurrent events (ICEs) for | |
| | analysis at Week 36 for the Primary Estimand | 31 |
| Table 4 | 4-3: Strategies for occurrence of intercurrent events (ICEs) for analysis at Week 3 | 6 for |
| | the Supplementary Estimand | |
| Table 4 | 4-4: Strategies for occurrence of intercurrent events (ICEs) for analysis at Week 3 | |
| | the Supplementary Estimand 2 | |
| Table 4 | 4-5: Shortening Criteria | 41 |


| Table 4-6: Strategies for occurrence of intercurrent events for analysis at week 64 for the | |
|---|---|
| Secondary Estimand | 42 |
| Table 4-7: Pre-defined laboratory abnormalities | 50 |
| Table 6-1: Pre-defined laboratory abnormalities | 60 |
| Table 6-2: PTs for selection of "Hypertension" | 61 |
| Table 6-3: PTs for selection of "Intraocular Inflammation" | 62 |
| Table 6-4: PTs for selection of "Nasal mucosal events" | |
| Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease" | 63 |
| Table 6-6: PTs for selection of medical history of "Ischaemic Heart Disease" | <b>70</b> |
| Table 6-7: PTs for selection of medical history of renal impairment requiring dialysis | 72 |
| Table 6-8: PTs for selection of medical history of "Hepatic Impairment" | 73 |
| Table 6-9: Recoding of NEI-VFQ 25 items | |
| Table 6-10: Sub-scales of the NEI-VFQ 25 score | 84 |
| Table 6-11: Strategies for displaying Summary Statistics in line with the primary estimand. | 85 |
| Table 6-12: Strategies for displaying Summary Statistic using imputation of missing values | |
| with LOCF | 86 |
| Table 6-13: Preliminary list of prohibited medication by drug names (may be updated before | ÷ |
| unmasking of the data) | 86 |
| Tables of Figures | |
| Figure 1–1: Study Design | 16 |
| Figure 1–2: Dosing Schedule | 17 |
| Figure 2–1: Hierarchical Hypothesis Testing | 20 |

# **Version History**

This Statistical Analysis Plan (SAP) for study 22153 is based on the protocol Version 1.0 dated 07 FEB 2023.

| SAP<br>Version | Date | Change | Rationale |
|---|---|---|---|
| 1 | 15 01<br>2024 | Not Applicable | Original version |
| 2 | 21 11<br>2024 | <ul> <li>Section 1.1: updated population attribute definition of both estimands.</li> <li>Section 1.1: updated table with inclusion of column including supplementary estimand 2</li> <li>Section 4.1: minor editorial updates</li> <li>Section 4.1.2.1: Handling of missing data and rules for imputing partial or missing start and end dates for medications and adverse events updated.</li> </ul> | More details<br>and<br>improvements<br>added;<br>Updates made<br>to align after |


- Section 4.1.3: Corrective stratification in analysis included to account for stratification errors and adjustments based on correct stratification categories, including the use of reading center data for RVO type

- Section 4.1.7: Minor edits made to the prohibited therapies list.
- Section 4.1.8: Update of the evaluation and classification of the imaging data, with specific rules for evaluating intraretinal fluid, subretinal fluid, retinal thickness, and fluorescein angiography assessments.
- Section 4.2.2: Added description that least-square mean change will be calculated with categorical covariates weighted as observed; minor updates to the description of the descriptive summary tables.
- Table 4.2 Updated to change days from +10 to +5.
- Section 4.2.3.1: Editorial updates in the description of the analysis as well as the SAS code; update of the estimation approach: single linear regression model including the treatment group variable with three levels instead of two pairwise regression models; added expression for the population-level summary.
- Section 4.3.2.: Minor edits for description of summary statistics.
- Section 4.3.2.1: Added clarification on handling the composite strategy for the ICE "premature discontinuation of study intervention due to treatment-related AEs," where the number of injections will be set to 9.
- Section 4.3.2.7: Updated the covariate description
- Section 4.3.2.8: Updated the statistical model used to account for the correct data collected.
- Sections 4.3.2.9/10/11: Minor editorial changes to reflects tables are provided already in Section 6.1.3.
- Section 4.3.2.12: Update definition for race subgroup analysis.
- Section 4.4: Minor editorial changes.
- Section 4.4.4: Added clarification regarding the exclusion of participants with no fluid at baseline, missing baseline information, or "undetermined" baseline fluid status from the analysis.
- Section 4.5.1: Minor editorial changes.
- Section 4.5.2.2: Minor editorial changes and removal of shift tables from the text.

review of TLF shells




- Section 4.6.2: Added clarification for pooling the two 8mg arms and updated the analysis for subgroup by RVO type to include descriptive summary statistics for additional secondary endpoints.
- Section 4.8: Added clarification about the change for the population attribute in the estimand definition from "participants" to "patients" for alignment with the target population
- Section 6.1: Minor editorial changes.
- Section 6.1.1: Minor editorial changes.
- Section 6.1.3.2: Minor editorial changes.
- Section 6.1.4: Removed the section on Kaplan-Meier analyses for time-to-treatment discontinuation and intake of prohibited medication and additional minor editorial changes
- Section 6.5: Minor editorial changes and removed the reference to the secondary estimand strategy and deleted the associated Table 6-13.
- Section 6.6: Added new section on identification of prohibited medication.


# **List of Abbreviations**

| Abbreviation | Description |
|--------------|-------------------------------------------------------------|
| ADE | adverse device effect |
| AE | adverse event |
| AESI | adverse events of special interest |
| ANCOVA | analysis of covariance |
| APAC | Asia-Pacific |
| APTC | anti-platelet trialists' collaboration |
| ATE | arterial thromboembolic events |
| AxMP | auxiliary medicinal product |
| BCVA | best-corrected visual acuity |
| BMI | body mass index |
| BRVO | branch retinal vein occlusion |
| CE | conformité européenne |
| CI | confidence interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CONSORT | Consolidated Standards of Reporting Trials |
| CRF | case report form |
| CRO | case report form contract research organization |
| CRVO | central retinal vein occlusion |
| CST | central subfield thickness |
| DL-AAA | |
| | DL-α-aminoadipic acid |
| DMC | data monitoring committee |
| DME | diabetic macular edema |
| DRM | dose regimen modification |
| eCRF | electronic case report form |
| ECG | electrocardiogram |
| EoS | end of study |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| EU | European Union |
| FA | fluorescein angiography |
| FAS | Full analysis set |
| FBR | future biomedical research |
| FDA | Food and Drug Administration |
| FP | fundus photography |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practice |
| HbA1c | hemoglobin A1c |
| HIPAA | Health Insurance Portability and Accountability Act |
| HRT | hormonal replacement therapy |
| HRVO | hemiretinal vein occlusion |
| IB | Investigator's Brochure |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug |
| IOP | intraocular pressure |
| IRF | intraretinal fluid |
| IRB | Institutional Review Board |
| IRT | Interactive Response Technology |
| IUD | intrauterine device |
| IUS | intrauterine hormone releasing system |
| IVT | Intravitreal(ly) |


| Abbreviation | Description |
|--------------|------------------------------------------------------------|
| LLOQ | Lower Limit of Quantification |
| MAR | Missing at Random |
| MDR | Medical Device Regulation |
| MMRM | mixed model for repeated measurements |
| nAMD | neovascular age-related macular degeneration |
| NEI-VFQ-25 | National Eye Institute Visual Functioning Questionnaire-25 |
| NI | non-inferiority |
| NVD | Neovascularization of the optic disc |
| OCT | optical coherence tomography |
| OCT-A | optical coherence tomography angiography |
| PCR | polymerase chain reaction |
| PCSV | potentially clinically significant value |
| PIGF | placental growth factor |
| PK | Pharmacokinetic |
| PKS | Pharmacokinetic analysis set |
| PT | preferred term |
| QoL | quality of life |
| Q4W | every 4 weeks |
| Q8W | every 8 weeks |
| RVO | retinal vein occlusion |
| SADE | serious adverse device effects |
| SAE | serious adverse event |
| SAF | Safety analysis set |
| SAP | statistical analysis plan |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SD-OCT | spectral domain optical coherence tomography |
| SDLL | Source Data Location List |
| SoA | schedule of activities |
| SOC | system organ class |
| SRF | sub-retinal fluid |
| SUSAR | suspected unexpected serious adverse reactions |
| T&E | treat and extend |
| TEAE | treatment-emergent adverse event |
| TMF | trial master file |
| ULOQ | Upper Limit of Quantification |
| US | United States |
| USPI | United States Prescribing Information |
| VEGF | vascular endothelial growth factor |
| VEGFR | vascular endothelial growth factor receptor |
| WOCBP | woman (women) of childbearing potential |
| YAG | yttrium-aluminum-garnet |


## 1. Introduction

Retinal vein occlusion (RVO) is one of the most frequent causes of visual loss from diseases affecting the retinal vessels of the eye (Rogers 2010). The 2 major RVO categories are central RVO (CRVO), with blockage of the single, central vein draining blood from the retina, and branch RVO (BRVO), where one or more of the branches of the central retinal vein are occluded. A less frequent subtype is hemiretinal vein occlusion (HRVO), where branches from the superior or inferior hemisphere are occluded, sharing characteristics with both CRVO and BRVO. RVO results in impaired venous drainage from the eye and retinal non-perfusion, leading to increased vascular endothelial growth factor (VEGF) expression. High VEGF levels can lead to macular edema, retinal hemorrhage, and neovascularization. Patients with central macular edema secondary to RVO lose visual acuity, and the visual prognosis, if untreated, is often poor (Holz 2013).

Intravitreal (IVT) anti-VEGF agents, including aflibercept 2 mg, have become the standard of care for the treatment of macular edema secondary to RVO, with a recommended dose of once every 4 weeks (Q4W). The goal of the current study is to test a IVT formulation with a higher concentration of aflibercept, aiming to increase the total amount of anti-VEGF therapeutic protein administered. This increased concentration has the potential to increase the drug's biological duration of action and provide greater efficacy. Additionally, it could reduce patient burden by extending the interval between IVT injections and reducing the overall number of doses. This reduction in treatment burden is particularly important for this population, many of whom are still working (United States Prescribing Information - USPI). The development candidate, aflibercept 8 mg (with a concentration of 114.3 mg/mL), targets IVT delivery of increased molar concentrations of VEGF inhibitors relative to the formulation currently approved for Eylea® 2 mg (USPI).

Aflibercept 8 mg has been proven to be effective and safe in adult patients with DME and nAMD in Phase 2/3 PHOTON and Phase 3 PULSAR studies, respectively. In DME, 91% to 89% of patients were able to maintain 12-16 week treatment intervals with the 8 mg formulation while achieving similar visual acuity results as the 2 mg formulation through Week 48. In nAMD, 79% to 77% of patients were able to maintain 12-16 week treatment intervals with the 8 mg formulation and achieved similar visual acuity results as the 2 mg formulation through Week 48. The safety profile of aflibercept 8 mg in both studies was consistent with the known safety profile of aflibercept 2 mg and no new safety signals were observed.

Study 22153 will investigate the efficacy and safety of aflibercept 8 mg in patients with RVO with the intent of achieving non-inferior BCVA gains from baseline, while extending the dosing interval to reduce the number of injections and potentially improving visual and/or anatomic outcomes for aflibercept 8 mg vs. the currently approved aflibercept 2 mg dose regimen as well as maintaining the same safety profile as aflibercept 2 mg.

This Statistical Analysis Plan (SAP) outlines the specific details of the required statistical analyses to be conducted at Week 36 and at Week 64, which corresponds to the end-of-study (EOS). No interim statistical analysis in the sense of a group-sequential or adaptive design will be performed. However, once all participants have completed Week 36 or discontinued prematurely, an analysis of all available data up to and including Week 36, including the primary estimand analysis, will be conducted using the database that has been locked after all subjects have completed the Week 36 visit (or discontinued). Subsequently, a final analysis of


all data, including the secondary estimand analysis, will be conducted after all participants have completed the study at Week 64 (or prematurely discontinued). The Week 36 endpoints will not be formally re-analyzed at the timepoint of the Week 64 analysis. The summary tables, figures, and listings (TFLs) that will be included in the Clinical Study Report (CSR) will be defined in a separate document. This SAP is based on the clinical study protocol version 1.0, dated February 7, 2023. All references to the study protocol henceforth refer to that version of the protocol.

# 1.1 Objectives, Endpoints, and Estimands

Table 1-1: Objectives and endpoints

| Ob | jectives | Endpoints |
|---|---|---|
| • | mary objective: To determine if treatment with aflibercept 8 mg Q8W provides non-inferior BCVA change compared to aflibercept 2 mg Q4W | Primary Endpoint: Change from baseline in BCVA measured by the ETDRS letter score at Week 36 |
| | condary objectives – Efficacy | |
| • | To determine if treatment with aflibercept 8 mg Q8W requires less injections compared to aflibercept 2 mg Q4W | <ul> <li>Key Secondary Endpoint</li> <li>Number of active injections from baseline to Week 64<sup>1</sup></li> <li>Secondary Endpoint</li> <li>Number of active injections from baseline to Week 36</li> </ul> |
| • | To determine the effect of aflibercept 8 mg Q8W compared to aflibercept 2 mg Q4W on other visual and anatomic measures of response | <ul> <li>Change from baseline in BCVA measured by the ETDRS letter score at Week 44²</li> <li>Change from baseline in BCVA measured by the ETDRS letter score at Week 64</li> <li>Participant gaining at least 15 letters in BCVA from baseline at Weeks 36 and 64</li> <li>Participant achieving an ETDRS letter score of at least 69 (approximate 20/40 Snellen equivalent) at Weeks 36 and 64</li> <li>Participant having no IRF and no SRF in the center subfield at Weeks 36 and 64</li> <li>Change from baseline in CST at Weeks 36 and 64</li> </ul> |
| • | To assess the efficacy of aflibercept 8 mg<br>Q8W compared to aflibercept 2 mg<br>aflibercept Q4W on vision-related QoL | Change from baseline in NEI-VFQ-25 total<br>score at Weeks 36 and 64 |
| Se | condary objective - Safety | |
| • | To evaluate the safety of aflibercept 8 mg<br>Q8W compared to aflibercept 2 mg<br>aflibercept Q4W | <ul> <li>Occurrence of TEAEs and SAEs through<br/>Weeks 36 and 64</li> </ul> |
| Se | condary objectives - Other | |
| • | To evaluate duration of effect of aflibercept 8 mg Q8W compared to aflibercept 2 mg aflibercept Q4W | <ul> <li>Participants dosed only Q8W through Week 36 in the 8 mg Q8W group</li> <li>Participant having last treatment interval ≥12 or of 16 weeks at Week 64</li> <li>Participant having next intended interval ≥12, ≥16 or of 20 weeks at Week 64</li> </ul> |


| Objectives | Endpoints |
|---|---|
| To evaluate the PK of aflibercept 8 mg Q8W compared to aflibercept 2 mg aflibercept Q4W | <ul> <li>Systemic exposure to aflibercept as<br/>assessed by plasma concentrations of free,<br/>adjusted bound and total aflibercept from<br/>baseline through Weeks 36 and 64</li> </ul> |
| Exploratory objectives | |
| To determine the effect of aflibercept 8 mg<br>Q8W compared to aflibercept 2 mg Q4W<br>on further visual and anatomic measures of<br>response | <ul> <li>Change from baseline in BCVA measured by the ETDRS letter score at each visit</li> <li>Participant with vision changes of at least 5, 10, or 15 letters in BCVA from baseline at each visit</li> <li>Participant with no IRF and no SRF in the center subfield at each visit</li> <li>Time to fluid-free retina over 36 and 64 weeks (total fluid, IRF, and/or SRF in the center subfield)</li> <li>Participant having sustained fluid-free retina over 36 and 64 weeks (total fluid, IRF, and/or SRF in the center subfield)</li> <li>Change in area of retinal ischemia at Weeks 36 and 64</li> <li>Change in the area of fluorescein leakage at Weeks 36 and 64</li> </ul> |
| To study molecular drivers of RVO or<br>related diseases, clinical efficacy of<br>aflibercept, and affected molecular<br>pathways | <ul> <li>Evaluation of clinical efficacy parameters by repertoire or frequency of genetic alterations (genomics substudy)</li> <li>Treatment related changes in circulating biomarkers (FBR)</li> </ul> |

AE=adverse event, BCVA=best-corrected visual acuity, CST=central subfield thickness, ETDRS=early treatment diabetic retinopathy study, FBR=future biomedical research, IRF=intraretinal fluid, NEI-VFQ-25=National Eye Institute Visual Functioning Questionnaire-25, PK=pharmacokinetics, QoL=quality of life, Q4W=every 4 weeks, Q8W=every 8 weeks, RVO=retinal vein occlusion, SAE=serious adverse event, SRF=sub-retinal fluid, TEAE=treatment-emergent adverse event

#### **Primary Estimand**

The primary estimand for the primary objective is described by the following attributes:

- Population: Adult patients with treatment-naïve macular edema secondary to RVO
- Endpoint: Change from baseline in BCVA measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score at Week 36
- Treatment condition:
  - Aflibercept 8 mg administered with 3 initial every 4 weeks (Q4W) initiation doses followed by extension of treatment interval to 8-weeks and further adjustment of intervals according to treatment response (8mg/3)
  - Aflibercept 8 mg administered with 5 initial Q4W initiation doses followed by extension of treatment interval to 8-weeks and further adjustment of intervals according to treatment response (8mg/5)
  - o Aflibercept 2 mg administered Q4W until Week 32, followed by adjustment of treatment intervals according to treatment response (2mg)

<sup>&</sup>lt;sup>1</sup> Where premature treatment discontinue due to treatment related AE is considered as treatment-failure and the number of active injections from baseline to Week 64 is set to an unfavorable outcome (equal to 16, the maximum value).

<sup>&</sup>lt;sup>2</sup> For the 8mg/5 and 2 mg groups only.


A delayed active injection resulting in an injection interval up to 4 weeks longer than planned is considered to be in line with the treatment regimen of interest.

- Intercurrent events and strategies:
  - Premature treatment discontinuation addressed by the hypothetical strategy (had participants continued treatment until Week 36)
  - Use of prohibited medication addressed by the hypothetical strategy (had prohibited medications not been taken)
  - Missed study intervention:
    - Missed active injection resulting in an injection interval up to 4 weeks longer than planned: treatment policy strategy (the effect of a missed active injection will be included in the estimate of the treatment effect)
    - Missed active injection resulting in an injection interval more than 4 weeks longer than planned: hypothetical strategy (had injection not been missed or delayed by less than 4 weeks)
- Population-level summary: Difference in mean change from baseline to Week 36 in BCVA between each aflibercept 8 mg group and the aflibercept 2 mg group

Rationale for estimand: A hypothetical strategy is mainly used to address intercurrent events (especially premature treatment discontinuation) since the aim is to show non-inferiority (NI) of aflibercept 8 mg vs. aflibercept 2 mg and using a hypothetical strategy would be a conservative approach since it prevents the treatment arms from appearing more similar. See Table 4-2 for details on the analysis approach for hypothetical strategy. For the intercurrent event "missed study intervention", a missed sham injection has no impact on the endpoint as no active treatment was missed and thus it is not considered as additional intercurrent event. The impact of other potential intercurrent events is expected to be negligible.

#### Supplementary Estimand for the primary estimand.

The supplementary estimands for the primary objective is defined in Table 1-2 in addition to the primary estimand.


Table 1-2: Supplementary Estimand for the Primary Objective

| | Primary Estimand | Supplementary Estimand 1 | Supplementary Estimand 2 |
|---|---|---|---|
| Population | Adult patients with treatment-naïve macular edema secondary to RVO. | Same as primary | Same as primary |
| Treatment condition | Aflibercept 8 mg administered with 3 initial every 4 weeks (Q4W) initiation doses followed by extension of treatment interval to 8-weeks and further adjustment of intervals according to treatment response Aflibercept 8 mg administered with 5 initial Q4W | Same as primary | Same as primary |
| | Aflibercept 8 mg administered with 5 initial Q4W initiation doses followed by extension of treatment interval to 8-weeks and further adjustment of intervals according to treatment response | | |
| | Aflibercept 2 mg administered Q4W until Week 32, followed by adjustment of treatment intervals according to treatment response | | |
| Variable<br>(endpoint) | Change from baseline in BCVA measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score at Week 36 | Same as primary | Same as primary |
| Population-level summary | Difference in mean change from baseline to Week 36 in BCVA between each aflibercept 8 mg group and the aflibercept 2 mg group | Same as primary | Same as primary |
| Intercurrent<br>events and<br>strategies | Premature treatment discontinuation – addressed<br>by the <u>hypothetical strategy</u> (had participants<br>continued treatment until Week 36) | Premature treatment<br>discontinuation – addressed by<br>the <u>treatment policy strategy</u><br>(the estimated treatment effect) | Premature treatment discontinuation Due to death: composite strategy (treatment) |

ersion 2.0 

| Primary Estimand | Supplementary Estimand 1 | Supplementary Estimand 2 |
|---|---|---|
| Primary Estimand Use of prohibited medication – address hypothetical strategy (had prohibited monot been taken) Missed study intervention: Missed active injection resulting in injection interval up to 4 weeks lon planned: treatment policy strategy of a missed active injection will be the estimate of the treatment effective. | supplementary Estimand 1 ed by the edications will consider the impact of early discontinuation of treatment) • Use of prohibited medication – addressed by the treatment policy strategy (effect of prohibited medications will be included in the estimate of the treatment effect) | Supplementary Estimand 2 discontinuation due to death is indicative of non-response) For any other reason that death: treatment policy strategy Use of prohibited medication addressed by the composite strategy (intake of prohibited |
| Missed active injection resulting in injection interval more than 4 week than planned: hypothetical strategy injection not been missed or delays than 4 weeks) | s longer o Missed active injection<br>y (had resulting in an injection | medication is indicative of non response) • Missed study intervention: ○ Same as Supplementary Estimand 1 |


## **Secondary Estimand**

The secondary estimand for the secondary objective "To determine if treatment with aflibercept 8 mg Q8W requires less injections compared to aflibercept 2 mg Q4W" is described by the following attributes:

- Population: Adult patients with treatment-naïve macular edema secondary to RVO
- Endpoint: Number of active injections from baseline to Week 64 where premature treatment discontinuations due to treatment related AE is considered as treatment-failure and the number of injections is set to an unfavorable outcome (equal to 16, the maximum value)
- Treatment condition:
  - Aflibercept 8 mg administered with 3 initial Q4W initiation doses followed by extension of treatment interval to 8-weeks and further adjustment of intervals according to treatment response
  - Aflibercept 8 mg administered with 5 initial Q4W initiation doses followed by extension of treatment interval to 8-weeks and further adjustment of intervals according to treatment response
  - Aflibercept 2 mg administered Q4W until Week 32, followed by adjustment of treatment intervals according to treatment response

The minimum treatment interval is 4 weeks while the study duration allows the maximum treatment interval to be 16 weeks. Imperfect adherence other than premature treatment discontinuation is considered as part of the treatment.

- Intercurrent events and strategies:
  - Premature treatment discontinuation
    - ➤ Due to lack-of-efficacy: Hypothetical strategy (had participants continued treatment until Week 64)
    - ➤ Due to treatment related AEs: Composite strategy (addressed in the endpoint definition)
    - ➤ Due to treatment unrelated AEs and other reasons: Hypothetical strategy (had participants continued treatment until Week 64)
  - Missed study intervention addressed by treatment policy strategy (the effect of a missed active injection will be included in the estimate of the treatment effect)
- Population-level summary: Difference in mean number of active injections up to Week 64 between each aflibercept 8 mg group and the aflibercept 2 mg group

Rationale for estimand: Premature discontinuation due to treatment related AE; usually these participants would stop treatment. However, this would make it appear as if these participants had a reduced burden with respect to the number of injections. To mitigate this and to assign a penalty (since this is regarded as treatment failure) an unfavorable outcome equal to the maximum possible (i.e., 16 injections) is assigned using the composite strategy. Premature discontinuation due to lack-of-efficacy is handled by the hypothetical strategy , as describe in Section 4.3.1.3, assuming that these participants would have continued study treatment with the maximum number of active injections possible with shortening of treatment interval in 4-week decrements (i.e., assuming they would meet the dose regimen modification (DRM) criteria for shortening at every dosing visit. For treatment unrelated AEs it is assumed that those participants could have continued in the study otherwise and behave similar to other


participants in the study arm and hence addressed by the hypothetical strategy. Missed study intervention is regarded as part of clinical practice and hence addressed by the treatment policy strategy. The impact of other potential intercurrent events is expected to be negligible.

## 1.2 Study Design

As show in Figure 1–1, this is a Phase 3, multi-center, randomized, double-masked, active-controlled clinical study to assess the efficacy and safety of high dose (8 mg) aflibercept compared to 2 mg aflibercept (both administered IVT) in participants with treatment-naïve macular edema secondary to RVO.

Figure 1-1: Study Design



BCVA=Best-corrected Visual Acuity, ETDRS=Early Treatment of Diabetic Retinopathy Study, NI=non-inferiority, Q4W=every 4 weeks, Q8W=every 8 weeks, RVO=retinal vein occlusion, T&E=treat and extend

Participants will be randomized in a 1:1:1 ratio to:

- Aflibercept 8 mg every 8 weeks (Q8W) after 3 initial Q4W initiation doses group (8 mg/3)
- Aflibercept 8 mg Q8W after 5 initial Q4W initiation doses group (8 mg/5)
- Aflibercept 2 mg Q4W group (2 mg)

The study consists of a screening/baseline period, a treatment period with a duration of 60 weeks, and an end of study (EoS) visit at Week 64. Details of the dosing schedule are shown in Figure 1–2. No study intervention will be administered at the end of study visit at Week 64.

The primary analysis will be performed at Week 36 once all participants have either completed this timepoint or discontinued prematurely. This analysis will not be repeated at Week 64. The final analysis will be conducted at Week 64, once all participants have either completed the study or discontinued prematurely. The analysis of the Week 36 efficacy endpoints will not be repeated at Week 64. The databases and analyses at Week 36 will only include study intervention information up to the visit prior to Week 36. For the Week 36


analysis, only data assessed prior to the study intervention will be part of the database/analyses. Further details are provided in a separate document "Data Cut-Off Specifications".

Figure 1-2: Dosing Schedule

| Year 1 | Day<br>1 | <u>Wk</u> 4 | <u>Wk</u> 8 | <u>Wk</u><br>12 | <u>Wk</u><br>16 | <u>Wk</u><br>20 | <u>Wk</u><br>24 | <u>Wk</u><br>28 | <u>Wk</u><br>32 | Wk<br>36<br>PE | <u>Wk</u><br>40 | Wk 44<br>SE <sup>1</sup> | <u>Wk</u><br>48 | <u>Wk</u><br>52 | <u>Wk</u><br>56 | <u>Wk</u><br>60 | Wk<br>64<br>KSE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| AFL 2 mg | Х | Х | Х | Х | Х | Х | Х | Х | Х | T&E | | | | | | - | |
| AFL 8 mg/3 | Х | Х | Х | 0 | Х | O <sup>2</sup> | Х | O <sup>2</sup> | Х | T&E- | | | | | | - | |
| AFL 8 mg/5 | Х | Х | Х | Х | X | 0 | Х | O <sup>2</sup> | Х | O <sup>2</sup> | Х | T&E | | | | | |
| | Shorte | ning C | riteria | : | | | | | Ex | tension | n Crite | Criteria: | | | | | |
| DRM | | VA los | | | | | , | | • | | | <5 letters | | | | • | ) |
| Criteria | >50 μm increase in CST from reference visit | | | | | | | ║. | CST thickness <320 µm including Bruch's<br>membrane / <300 µm excluding Bruch's membrane | | | | | | | brane | |
| | Interval shortening possible from W16 for 8 mg/3, W24 for 8 mg/5, and W40 for 2mg | | | | | | | | - 11 | Interval extension possible from W32 for 8 mg/3, W40 for 8 mg/5 and W32 for 2 mg | | | | | | N40 | |
| | Refere | Reference is W12 for 8 mg/3, W20 for 8 mg/5 and 2 mg | | | | | | | | | is W | 12 for 8 ı | mg/3, | W20 f | or 8 mg | g/5 and | l 2 mg |

AFL=aflibercept, BCVA=best-corrected visual acuity, CST=central subfield thickness, DRM=dose regimen modification, KSE=key secondary endpoint, O=sham injection visit, PE=primary endpoint, SE=secondary endpoint, SD-OCT=spectral domain optical coherence tomography, T&E=treat and extend, Wk=week, X=active injection visit, -=no injection, 8 mg/3=8 mg Q8W after 3 initial Q4W doses, 8 mg/5=8 mg Q8W after 5 initial Q4W doses.

<sup>1</sup>=Secondary endpoint BCVA change from baseline to Week 44 for 2 mg and 8 mg/5 groups.

<sup>&</sup>lt;sup>2</sup>=Participants meeting interval shortening criteria at any dosing visit starting from Week 16 for 8 mg/3, Week 24 for 8 mg/5 or Week 40 for 2 mg have their dosing interval shortened by 4 weeks. Interval extension is possible from Week 32 for 8 mg/3, from Week 40 for 8 mg/5, and from Week 32 for 2 mg depending on DRM.


# 2. Statistical Hypotheses

The one-sided test hypotheses in relation to the primary and two-sided test hypotheses in relation to the secondary estimands, are described according to the fixed hierarchical order planned for their testing.

1. The first test problem (related to the primary estimand) involves the non-inferiority testing of 8 mg 5 loads vs 2mg:

Null hypothesis  $H_{01}$ :  $\mu_{1.5} \le \mu_0 - 4$  vs. alternative hypothesis  $H_{11}$ :  $\mu_{1.5} > \mu_0 - 4$ 

Where  $\mu_{1.5}$  and  $\mu_0$  represent the group means for the change from baseline in BCVA at Week 36 for the 8 mg/5 group and the 2 mg group, respectively.

Note that larger values measured for the change from baseline in BCVA are better. The aim is to show that the 8 mg/5 group is no less effective than the existing the 2 mg group, using a NI margin of 4 letters for the difference of the means.

2. The second test problem (related to the primary estimand) involves the non-inferiority testing of 8 mg 3 loads vs 2mg:

Null hypothesis  $H_{02}$ :  $\mu_{1.3} \le \mu_0 - 4$  vs. alternative hypothesis  $H_{12}$ :  $\mu_{1.3} > \mu_0 - 4$ 

Where  $\mu_{1.3}$  and  $\mu_0$  represent the group means for the change from baseline in BCVA at Week 36 for the 8 mg/3 group and the 2 mg group, respectively.

Note that larger values measured for the change from baseline in BCVA are better. The aim is to show that the 8 mg/3 group is no less effective than the existing the 2 mg group, using a NI margin of 4 letters for the difference of the means.

3. The third test problem (related to the secondary estimand) focuses on comparing the conditional distributions for the number of active injections between the 8 mg 3 loads and 2 mg groups:

Null hypothesis  $H_{03}$ :  $f_3(Y_1|X) = g(Y_2|X)$  vs. alternative hypothesis  $H_{13}$ :  $f_3(Y_1|X) \neq g(Y_2|X)$ 

Where  $f_3(Y_1|X)$  and  $g(Y_2|X)$  represent the conditional distributions for the number of active injections Y conditional on the data X from baseline to Week 64 for the 8 mg/3 group and the 2 mg group, respectively.

Note that smaller values for the number of active injections are better. The aim is to show that the 8 mg/3 group is superior to the existing the 2 mg group in that it leads to fewer injections. Thus, the null hypothesis should be rejected in favor of the alternative hypothesis and the estimate of the treatment effect based on a linear regression model adjusted for the stratification variables should favor the 8 mg/3 group.

4. The fourth test problem (related to the secondary estimand) focuses on comparing the conditional distributions for the number of active injections between the 8 mg 5 loads and 2 mg groups:

Null hypothesis  $H_{04}$ :  $f_5(Y_1|X) = g(Y_2|X)$  vs. alternative hypothesis  $H_{14}$ :  $f_5(Y_1|X) \neq g(Y_2|X)$ 

Where  $f_5(Y_1|X)$  and  $g(Y_2|X)$  represent the conditional distributions for the number of active injections Y conditional on the data X from baseline to Week 64 for the 8 mg/5 group and the 2 mg group, respectively.


Note that smaller values for the number of active injections are better. The aim is to show that the 8 mg/5 group is superior to the existing the 2 mg group in that it leads to fewer injections. Thus, the null hypothesis should be rejected in favor of the alternative hypothesis and the estimate of the treatment effect based on a linear regression model adjusted for the stratification variables should favor the 8 mg/5 group.

5. The fifth test problem (related to the primary estimand) involves the superiority testing of 8 mg 5 loads vs 2mg:

Null hypothesis  $H_{05}$ :  $\mu_{1.5} \le \mu_0$  vs. alternative hypothesis  $H_{15}$ :  $\mu_{1.5} > \mu_0$ 

Where  $\mu_{1.5}$  and  $\mu_0$  represent the group means for the change from baseline in BCVA at Week 36 for the 8 mg/5 group and the 2 mg group, respectively.

Note that larger values measured for the change from baseline in BCVA are better. The aim is to show that the 8 mg/5 group is superior to the existing the 2 mg group.

6. The sixth test problem (related to the primary estimand) involves the superiority testing of 8 mg 3 loads vs 2mg:

Null hypothesis  $H_{06}$ :  $\mu_{1.3} \le \mu_0$  vs. alternative hypothesis  $H_{16}$ :  $\mu_{1.3} > \mu_0$ 

Where  $\mu_{1.3}$  and  $\mu_0$  represent the group means for the change from baseline in BCVA at Week 36 for the 8 mg/3 group and the 2 mg group, respectively.

Note that larger values measured for the change from baseline in BCVA are better. The aim is to show that the 8 mg/3 group is superior to the existing the 2 mg group.

Justification for the NI margin can be found in Section 9.1 of the study protocol.

## 2.1 Multiplicity Adjustment

As shown in Figure 2–1 and described in Section 2 a hierarchical testing procedure will be used to control the overall family-wise type I error in the strong sense. The statistical comparisons will be carried out in the hierarchical order as defined for the hypotheses in Section 2. Consequently, the second, third, fourth, fifth, and sixth null hypotheses will only be tested if the previous comparisons were in favor of the 8 mg/5 group or 8 mg/3 group in that the previous null hypotheses were rejected and, for two-sided null hypotheses only, the related estimate supported a superiority of the corresponding 8 mg arm. Operationally the non-inferiority and superiority hypotheses will be evaluated by one-sided tests with a significance level of 0.025, and the hypotheses for comparing number of active injections will be evaluated by two-sided tests with a significance level of 0.05. Two-sided 95% CIs for the treatment difference will be reported corresponding to all hypotheses.




Figure 2-1: Hierarchical Hypothesis Testing

8/5 BCVA36 = Group means for the change from baseline in BCVA at Week 36 for the 8 mg/5 group and the 2 mg group. Testing Non-inferiority of 8 mg/5 vs 2mg.

8/3 BCVA36 = Group means for the change from baseline in BCVA at Week 36 for the 8 mg/3 group and the 2 mg group. Testing Non-inferiority of 8 mg/3 vs 2mg.

8/3 Numlnj64= Conditional distributions for the number of active injections from baseline to Week 64 for the 8 mg/3 group and the 2 mg group.

8/5 Numlnj64= Conditional distributions for the number of active injections from baseline to Week 64 for the 8 mg/5 group and the 2 mg group.

8/5 BCVA36 Sup= Group means for the change from baseline in BCVA at Week 36 for the 8 mg/5 group and the 2 mg group. Testing Superiority of 8 mg/5 vs 2mg.

8/3 BCVA36 Sup= Group means for the change from baseline in BCVA at Week 36 for the 8 mg/3 group and the 2 mg group. Testing Superiority of 8 mg/3 vs 2mg.


# 3. Analysis Sets

For the purpose of analysis, the following analysis sets are defined:

Table 3-1: Analysis Sets

| Participant Analysis Set | Description |
|---|---|
| Full analysis set (FAS) | All participants randomly assigned to study intervention who were exposed to study intervention at least once. |
| Safety analysis set (SAF) | All participants randomly assigned to study intervention who were exposed to study intervention at least once. |
| Pharmacokinetic analysis set (PKS) | All participants randomly assigned to study intervention with at least one non missing PK result after the first dose of study intervention. |

PK=pharmacokinetic

#### Full analysis set (FAS)

The Full Analysis Set (FAS) will consist of all participants who have been randomly assigned to the study intervention and who were exposed to study intervention at least once. The participants will be analyzed based on their original randomized group. This approach ensures that the analysis accurately reflects the participants' original randomization status, thereby maintaining the integrity of the study results. The FAS will be used to analyze endpoints related to efficacy.

#### Safety analysis set (SAF)

The Safety analysis set (SAF) will consist of all participants who have been randomly assigned to the study intervention and who have received at least one dose of the study intervention. The analysis of the SAF will be based on the actual treatment the participant received during the study (as treated). This means that the participant's exposure to the study intervention will be accounted for and considered in the analysis, regardless of any deviations from the planned intervention. The SAF will be used to analyze the endpoints and assessments related to safety.

## Pharmacokinetic analysis set (PKS)

The Pharmacokinetic analysis set (PKS) will consist of all participants who have been randomly assigned to study interventions and have recorded at least one non-missing PK measurement after the first dose of the study intervention. The analysis of the PKS will be based on the treatment that the participant actually received, not necessarily on the treatment that they were initially assigned to receive (as treated analysis).

#### As randomized versus as treated

The only systematic deviation from the randomized treatment that may occur is due to a systematic error in the IXRS system set up. Therefore, it is assumed that participants are generally treated as randomized, meaning the randomized treatment group is considered the actual treatment group, unless the participant did not receive any treatment after randomization. However, isolated instances of incorrect treatment at specific timepoints will not change the "as treated" assignment. Any participant whose "as treated" assignment differs from their "as randomized" assignment will be specifically listed.

Final decisions regarding the assignment of participants to analysis sets will be made during the review of study data and documented in the final list of important deviations, validity findings and assignment to analysis set(s).


# 4. Statistical Analyses

#### 4.1 General Considerations

The testing of the primary and secondary endpoints is performed at an overall significance level of 0.025 for one-sided tests and 0.05 for two-sided tests, along with reporting of two-sided 95% CIs for these tests. The testing strategy is defined in Section 2.1. For descriptive purposes of other endpoints, 95% two-sided CIs will be provided where applicable.

The summary of continuous data will include the number of observations, mean, standard deviation (SD), median, quartiles, minimum, and maximum.

For categorical data, the summary will include the number of participants who provided data at the relevant time point (n), frequency counts, and percentages. The percentages will be presented to one decimal place but will not be reported for zero counts. The calculation of percentages will use n (the number of observations with non-missing values) as the denominator, unless otherwise specified in the output.

Number of decimal places for summary statistics will be the following:

Statistic Number of digits Same as original data Minimum, maximum Mean, median 1 more than in original data 1 more than in original data SD Frequencies (%) 1 digit **Ouartiles** 1 more than in original data Confidence Intervals (CI) 1 more than in original data p-values 4 digits

Table 4-1: Number of decimal places for summary statistics

Additionally, where applicable, descriptive summary tables for efficacy endpoints will be provided by treatment group and visit for and based on:

- All observed cases regardless of the occurrence of an ICE in the FAS population
- All observed cases until the occurrence of an ICE in line with the primary estimand strategy in the FAS population (see Table 6-11 in Section 6.5),
- All observed cases until the occurrence of an ICE with imputation of missing values with LOCF in the FAS population (see Table 6-12 in Section 6.5)

The statistical evaluation will be performed by using the software SAS (release 9.4 or higher; SAS Institute Inc., Cary, NC, USA) and/or R (R Core Team 2013, R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL http://www.R-project.org/).

The exclusion of participants from the primary analysis will be determined during the Data Review Meeting (on masked data) that will be held in accordance with ICH E9 prior to the database freeze on Week 36 data. Only participants who have completed Week 36 will be included in the analysis.


# **4.1.1 Definition of Dropouts**

In the context of this study, dropouts will be defined as participants who withdraw or prematurely discontinue both their participation in the study and the study intervention, regardless of the reason. This definition also encompasses participants who are lost to follow-up, meaning their status cannot be determined or they are unable to be contacted. The primary reasons for withdrawing will be collected in the eCRF and tabulated accordingly.

# 4.1.2 Handling of Missing Data

All missing or incomplete data will be displayed in the participant data listing exactly as it is recorded in the eCRF.

#### 4.1.2.1 General Rules

The following rules will be applied where applicable to ensure that participants are not excluded from statistical analysis due to missing or incomplete data:

#### • Efficacy Variables

The statistical methods for handling missing data resulting from participant discontinuing the study will be dealt with in line with the corresponding estimand strategies and are outlined in Section 4.2.2 and in Section 4.3.1.2., as applicable.

#### Concomitant medication and adverse events

For Adverse Events (AEs) and prior/concomitant medications, complete start and stop dates must be recorded to determine if the AE occurred during the study intervention period (i.e. treatment-emergent) or the medication was taken during the study intervention period (i.e. concomitant). In case of partial dates, the following rules will be applied

For partial/missing start dates of medications and AEs, impute as follows to determine whether concomitant and treatment-emergent, respectively:

- If only the month and year of the start date is available and the end date is after (or unclear due to missingness) the date of the first study intervention:
  - o If the month/year of the start date equals the month/year of first study intervention, then impute as the date of first study intervention.
  - o If the month/year of the start date is before the month/year of first study intervention, then impute as the last day of that month/year.
  - o If the month/year of the start date is after the month/year of first study intervention, then impute as the first day of that month/year.
- If only the year of the start date is available, and the end date is after (or unclear due to missingness) the date of the first study intervention:
  - o If the year of the start date equals the year of first study intervention, then impute as the date of first study intervention.
  - o If the year of the start date is before the year of first study intervention, then impute as the last day and month of that year.
  - o If the year of the start date is after the year of first study intervention, then impute as the first day and month of that year.


• If the start date is entirely missing and the end date is after (or unclear due to missingness) the date of the first study intervention, then impute as the date of first study intervention.

For partial/missing end dates of medications, impute as follows to determine whether concomitant:

- If only the month and year of the end date is available, and the start date is before (or unclear due to missingness) the date of the last study intervention:
  - o If the month/year of the end date equals the month/year of last study intervention, then impute as the date of last study intervention.
  - o If the month/year of the end date is before the month/year of last study intervention, then impute as the last day of that month/year.
  - o If the month/year of the end date is after the month/year of last study intervention, then impute as the first day of that month/year.
- If only the year of the end date is available, and the start date is before (or unclear due to missingness) the date of the last study intervention:
  - o If the year of the end date equals the year of last study intervention, then impute as the date of last study intervention.
  - o If the year of the end date is before the year of last study intervention, then impute as the last day of that year.
  - o If the year of the end date is after the year of last study intervention, then impute as the first day of that year.
- If the end date is entirely missing and the start date is before (or unclear due to missingness) the date of the last study intervention, then impute as the date of last study intervention.

Imputed dates will only be used for summary tables. Original (partial) entries will be retained in listings.

#### 4.1.3 Data Rules

**Definition of baseline:** The latest available valid measurement at or before the start of study intervention will be used as baseline value for all assessments, unless specified otherwise. These measurements may be taken either at the screening visit (Visit 1) or the baseline visit (Visit 2), depending on the study's planned procedure timeline. The detailed timing of study procedures can be found in the study protocol.

For systolic and diastolic blood pressure, the baseline value is determined by averaging all of the measurements taken at or prior to randomization. It is important to note that any measurements taken during the initial screening visit will not be included in the calculation if the participant failed to meet the screening criteria.

**Change from baseline:** The absolute change from baseline will be calculated by subtracting the baseline value from the value obtained during treatment/follow-up. The formula for this calculation is:


Absolute Change = post-baseline value – baseline value.

Additionally, some parameters may also be analyzed as relative change, which is calculated as the percentage change from the baseline value. This calculation is defined as:

Relative change = 100 \* [(post-baseline value – baseline value) / baseline value].

**Laboratory values < LLOQ or > ULOQ :** For laboratory values which are given as < LLOQ, half the value of the LLOQ will be used for analysis. Differences between two values < LLOQ will be assigned values of 0, and ratios between two values < LLOQ will be assigned a value of 1. For PK values, those under < LLOQ will be set to LLOQ/2 for geometric mean statistics in PK analysis but set to 0 for arithmetic statistics (mean, SD, CV). For values > ULOQ, the value of ULOQ will be used for analysis.

Repeated measurements at the same visit after start of treatment: If more than one post-randomization measurement is available for a given visit, the first valid observation will be used in the data summaries and all observations will be presented in the data listings.

Corrective Stratification in Analysis: in the event of stratification errors with respect to the stratification variables (geographic region [Japan vs. APAC vs Europe vs America], categorized baseline BCVA [<60 vs. ≥60], and RVO type [CRVO/HRVO vs BRVO]) at the time of randomization, analyses will be conducted based on participants' correct stratification category. Additionally, for RVO type the category will be derived from the reading center data. In case of missing reading center data, the RVO type category based on the investigator assessment as used for the randomization will be used.

#### 4.1.4 Unscheduled Assessments

To provide an accurate representation of the data collected, measurements taken at unscheduled visits will be displayed in individual subject data listings. However, these measurements will not be incorporated into the general summary tables for the data. Should multiple measurements of the same variable be taken during an unscheduled visit, all the measurements will be displayed in the relevant subject data listing.

## 4.1.5 End of Study / Early Discontinuation Visit

Participants are allowed to discontinue the study intervention prematurely. This can happen at any point during the study. However, regardless of when the premature discontinuation occurs, all required assessments must be completed according to the protocol for the end-of-study (EOS) or early-discontinuation (ED) visit.

If participants discontinue study prematurely, the visit-based information recorded in the EOS/ED visit folder will be re-mapped to the relevant regular study visit, provided the EOS/ED visit falls within the appropriate visit window and the corresponding regular visit has not taken place. If any visit-based information cannot be re-mapped to a regular visit, it will be treated as an unscheduled assessment and managed accordingly as described in Section 4.1.4.

For participants who complete the study and intervention, no re-mapping is necessary, but the visit-based information in the EOS/ED visit folder will be assigned to "Week 64" and presented in the summary tables as such.


It is important to note that for some variables, data may be collected at visits where this variable was not scheduled to be collected. However, this data will still be used in last observation carried forward (LOCF) analyses when applicable. Descriptive by-visit summary tables and repeated measurement analyses should only include data from pre-planned, visits for which the respective variable was scheduled to be collected.

# Mapping of selected assessments to regular study visits

The following assessments will be mapped:

- BCVA (ETDRS) and Refraction
- IOP
- Slit Lamp Examination
- Indirect Ophthalmoscopy
- SD-OCT
- Vital signs
- Pregnancy test

The following rule will be used:

• If EOS/ED visit performed within visit window of a regular study visit (as specified in the "Schedule of Activities" in the protocol), then re-mapping to regular study visit

For example, if a participant discontinued prematurely (study and/or study intervention) at the timing of Visit 3 / Week 4 (i.e. EOS/ED visit date = study day 29±5 days), then any of the assessments listed above recorded in the EOS/ED visit folder will be re-mapped to regular study Visit 3, unless a regular study Visit 3 was already performed.

#### 4.1.6 Definition of Fellow-Eve Treatment

The treatment of the fellow eye will be documented on the Concomitant Medication page in the eCRF by specifying the fellow eye that was treated.

Any medication given prior to the first dose of the study intervention will be considered prior treatment for the fellow eye, while any medication given after the first dose of the study intervention will be considered concomitant bilateral treatment. The rules for partially missing dates will apply as described in section 4.1.2.1.

#### 4.1.7 Definition of Prohibited Medications

The following medications are prohibited, as identified on the prior and concomitant medication page:

- Any of the following anti-VEGF medications administered in the study eye:
  - o Aflibercept (trade name: Eylea), unless administered as study intervention
  - Bevacizumab (trade name: Avastin)
  - o Brolucizumab (trade name: Beovu)
  - Ranibizumab (trade name: Lucentis)
  - o Faricimab (trade name: Vabysmo)


- o Conbercept (trade name Lumitin)
- o Pegaptanib sodium (trade name: Macugen)
- Treatment with intraocular or periocular implant in the study eye.
- Administration of systemic anti-angiogenic medications for any condition.
- Use of intraocular or periocular steroids for the treatment of RVO, or steroid implants in the study eye.
- Treatment with ocriplasmin in the study eye.
- Gene therapy, or cell therapy in the study eye or fellow eye.

Additionally, the following surgical procedures are prohibited:

- Treatment with retinal laser photocoagulation for the treatment of RVO in the study eye.
- Treatment with vitrectomy surgery in the study eye.

The investigator may administer any medication that is deemed necessary for the participant's well-being and is not expected to affect the evaluation of the study intervention.

Both the prohibited medications and the prohibited procedures outlined above count towards the intercurrent event "Use of prohibited medication" that is used in the definition of the primary estimand (see Section 1.1).

Please refer to Section 6.6 on details how to identify intake of prohibited medications and cases of prohibited procedures during the study.

## 4.1.8 Imaging data assessed by the reading center

If imaging data have been assessed by the reading center, but were also captured in the eCRF, only the data assessed by the reading center will be used for the analysis unless otherwise stated.

In summary tables the following parameters will be evaluated and classified as follows:

From spectral domain optical coherence tomography (SD-OCT) assessment:

- Intraretinal fluid (IRF) in central subfield (Reading center variables: Intraretinal fluid (IRF: cystoid edema) present and IRF in the central 1mm affected):
  - $\circ$  IRF = No (if any of them is ticked):
    - IRF presence = No
    - IRF presence = Yes AND IRF in the central 1mm = No or QT
    - IRF presence = QT
  - $\circ$  IRF = Yes:
    - IRF presence = Yes AND IRF in the central 1mm = Yes
  - o IRF = Undetermined (if any of them is ticked):
    - IRF presence = CG


- IRF presence = Yes AND IRF in the central 1mm = CG
- Subretinal fluid (SRF) in <u>central subfield</u> (Reading center variables: Subretinal fluid (SRF) present and SRF in the central 1mm involved):
  - o SRF = No (if any of them is ticked):
    - SRF presence = No
    - SRF presence = Yes AND SRF in the central 1mm = No or QT
    - SRF presence = QT
  - $\circ$  SRF = Yes:
    - SRF presence = Yes AND SRF in the central 1mm = Yes
  - o SRF = Undetermined (if any of them is ticked):
    - SRF presence = CG
    - SRF presence = Yes AND SRF in the central 1mm = CG
- Central subfield thickness (CST)
  - o Retinal thickness in central subfield
    - o CST = reported value in  $\mu$ m
    - o If CG, set to missing

From fluorescein angiography (FA) assessment:

- Area of retinal ischemia (Reading center variables: 'Presence of perifoveal and parafoveal ischemia' and 'total area of macular ischemia (not considering the FAZ)')
  - o If Yes
    - Area = reported value in mm<sup>2</sup>
  - If No
    - Area = 0
  - If QT
    - Area = 0
  - o If CG
    - Set to missing
- Area of fluorescein leakage (Reading center variables: 'Presence of macular leakage' and 'area of macular leakage')
  - If Yes
    - Area = reported value in  $mm^2$
  - If No


- Area = 0
- If OT
  - Area = 0
- o If CG
  - Set to missing

# 4.2 Primary Endpoint Analysis

The testing of the primary and key secondary endpoints is performed at an overall significance level of 0.025 for the one-sided tests and 0.05 for the two-sided tests. The testing strategy is defined in Section 2.1. The 95% two-sided CIs will also be provided as applicable.

# **4.2.1 Definition of Endpoint**

The primary endpoint is the change from baseline in BCVA (as measured by ETDRS letter score) at Week 36.

# 4.2.2 Main Analytical Approach

For the primary analysis of the primary efficacy variable, a mixed model for repeated measurements (MMRM) will be used with baseline BCVA measurement as a covariate and treatment group (2q4 vs 8q8/3 vs 8q8/5), visit (up to Week 36), and the stratification variables (geographic region [Japan vs. APAC vs Europe vs America], categorized baseline BCVA [<60 vs. ≥60], and RVO type [CRVO/HRVO vs BRVO]) as fixed factors as well as terms for the interaction between baseline and visit (up to Week 36) and for the interaction between treatment and visit (up to Week 36). Only data up to Week 36 will be included for this analysis. A Kenward-Roger approximation will be used for the denominator degrees of freedom. Further, an unstructured covariance structure will be used to model the within-subject error, assuming different covariance parameters per treatment group. The unstructured covariance structure will be used since it avoids making any assumptions on the correlations between repeated measures. If the fit of the unstructured covariance structure fails to converge, the following covariance structures will be tried in order until convergence is reached: Toeplitz with heterogeneity, autoregressive with heterogeneity, Toeplitz, autoregressive and compound symmetry.

$$Y_{ijk} = \beta_0 + x_i \times \beta_{base} + \beta_{type}^{(t)} + \beta_{reg}^{(l)} + \beta_{base\_cat}^{(m)} + \beta_{treat}^{(k)} + \beta_{visit}^{(j)} + x_i \times \beta_{base*visit}^{(j)} + \beta_{treat*visit}^{(k,j)} + \epsilon_{ijk}$$

with

- $Y_{ijk}$  being the change from baseline to visit j for the participant i receiving treatment k
- $\beta_0$  being the intercept
- $x_i$  being the baseline BCVA measurement of participant i
- $\beta_{base}$  the fixed effect of the baseline BCVA measurement
- $\beta_{type}^{(t)}$  the fixed effect of RVO type t
- $\beta_{reg}^{(l)}$  the fixed effect of region 1 (as recorded on the eCRF),
- $\beta_{base\_cat}^{(m)}$  the fixed effect of categorized baseline BCVA measurement m


- $\beta_{treat}^{(k)}$  the fixed effect of treatment k
- $\beta_{visit}^{(j)}$  the fixed effect of visit j
- $\beta_{base*visit}^{(j)}$  the interaction between baseline BCVA and visit j
- $\beta_{treat*visit}^{(k,j)}$  the interaction between treatment k and visit j
- $\epsilon_{ijk}$  the residual error with  $\epsilon_{ijk} \sim N(0, \sigma_{jk}^2)$  and  $corr(\epsilon_{ijk}, \epsilon_{ij'k}) = \rho^k \{j, j'\}$

In terms of the model parameters the population-level summary for the primary estimand (i.e., the treatment effect at Week 36) can then be expressed as

$$D_{8/3} = \left[\beta_{treat}^{(8mg/3)} + \beta_{treat*visit}^{(8mg/3,w36)}\right] - \left[\beta_{treat}^{(2mg)} + \beta_{treat*visit}^{(2mg,w36)}\right]$$

for the comparison of 8mg/3 vs 2 mg and

$$D_{8/5} = \left[\beta_{treat}^{(8mg/5)} + \beta_{treat*visit}^{(8mg/5,w36)}\right] - \left[\beta_{treat}^{(2mg)} + \beta_{treat*visit}^{(2mg,w36)}\right]$$

for the comparison of 8mg/5 vs 2 mg.

The primary analysis will be conducted using the FAS. Participants will be analyzed within their original randomized intervention group, regardless of any modifications in their dose interval as per DRM criteria.

In accordance with the primary estimand and approach to intercurrent events of premature treatment discontinuation, no explicit imputation will be performed for missing BCVA measurements. Instead, missing BCVA measurements will be assumed to be missing at random (MAR) and will be handled by the MMRM model. This model will account for the missing data and provide a more robust estimate of the treatment effect.

Summary tables will include number of participants, least-square mean (LSmean) change (with categorical covariates weighted as observed), (unadjusted) mean change and SD and baseline means of each treatment group. For non-inferiority and superiority testing the estimates expressed as LSmean change, the test statistics, the degrees of freedom and corresponding p-values will be presented. Two-sided 95% confidence intervals will be provided as well.

An overview of the implementation strategies for handling of intercurrent events is described in Section 4.2.2.1.

Descriptive summary tables will be provided by treatment group and visit as described in Section 4.1 for:

- all observed cases regardless of the occurrence on an ICE,
- all observed cases until the occurrence of an ICE in line with the estimand strategy,
- all observed cases until the occurrence of an ICE with imputation of missing values using LOCF.

#### 4.2.2.1 Strategies for occurrence of intercurrent events

Analysis strategies for intercurrent events for the primary estimand occurring through Week 36 are described in Table 4-2 below.


Table 4-2: Implementation strategies for the handling of intercurrent events (ICEs) for analysis at Week 36 for the Primary Estimand

| ICE Strategies for the Primary Estimand | | | |
|---|---|---|---|
| Intercurrent event | Strategy | Main Analysis | Sensitivity Analysis |
| Premature<br>discontinuation of<br>study intervention<br>for any reason before<br>Week 36 | Hypothetical | and discontinuation of study: non-<br>observed data beyond<br>discontinuation of study intervention<br>will be covered implicitly in the<br>MMRM | Non-observed data beyond discontinuation of study intervention will be imputed by LOCF |
| | | and continuation of study: observed data beyond last active injection (that was administered before the premature discontinuation of study intervention) + current treatment interval +5 days will be excluded from analysis and resulting missing data will be covered implicitly in the MMRM | Observed data beyond last active injection (that was administered before the premature discontinuation of study intervention) + current treatment interval +5 days will be excluded from analysis and resulting missing data will be imputed by LOCF |
| Use of a prohibited medication (as per section 4.1.7) before Week 36 | Hypothetical | Observed data beyond first administration of the prohibited medication in study eye will be excluded from analysis and resulting missing data will be covered implicitly in the MMRM | Observed data beyond first administration of the prohibited medication in study eye will be gexcluded from analysis and resulting missing data will be imputed by LOCF |
| Missed active injection resulting in an actual injection interval up to 4 weeks longer than planned | Treatment policy | y All observed data will be <u>included</u> in<br>the analysis and the MMRM | All observed data will be <u>included</u> in the analysis |
| Missed active injection resulting in an actual injection interval more than 4 weeks longer than planned | Hypothetical | Observed data beyond last active injection (that was administered before the first missed active injection) + current treatment interva +5 days will be excluded from analysis and resulting missing data will be covered implicitly in the MMRM | Observed data beyond last active injection (that was administered before the first missed active dinjection) + current treatment interval +5 days will be excluded from analysis and resulting missing data will be imputed by LOCF |

# 4.2.3 Sensitivity Analyses

In addition to the MMRM approach described above, we will conduct three additional sensitivity analyses.

Firstly, we will use the Last Observation Carried Forward (LOCF) method until Week 36 to impute missing post-baseline BCVA values of participants who have at least one post-baseline value.

Secondly, we will apply Multiple Imputation (MI) assuming Missing at Random (MAR) to impute missing post-baseline BCVA values. For both LOCF and MI, we will use ANCOVA to analyze the change from baseline in BCVA at Week 36.


Thirdly, we will assess the sensitivity of the MI results in the second sensitivity analyses to deviations from the MAR assumption. To do this, we will conduct a tipping point analysis.

# 4.2.3.1 ANCOVA using LOCF

The sensitivity analysis of the primary efficacy endpoint using an ANCOVA with LOCF follows the same estimand strategy as the primary analysis. Observed data after occurrence of ICE will be handled as described in Table 4-2.

Baseline BCVA measurement will be included as a covariate, while treatment group (2q4 vs 8q8/3 vs 8q8/5) and stratification variables (geographic region [Japan vs. APAC vs Europe vs America], baseline BCVA [<60 vs. ≥60]), and RVO type ([CRVO or HRVO] vs BRVO) will be treated as fixed factors. Variance terms will be estimated separately for each of the three treatment groups.

The observation at Week 36 of participant i receiving treatment t can be written as follows:

$$Y_{itrb} = \mu_t + \gamma_r + \eta_b + \omega_p + x_i \beta + \epsilon_{itrb}$$

with

- $Y_{itrb}$  being the change from baseline to Week 36 for the ith participant,
- $\mu_t$  being the treatment effect,
- $\gamma_r$  being the geographic region effect (as recorded on the eCRF),
- $\eta_b$  being the categorical baseline BCVA (<60 vs.  $\geq$ 60; as recorded on the eCRF),
- $\omega_p$  being the RVO type effect,
- $x_i$  being the baseline BCVA measurement of participant i,
- $\epsilon_{itrb}$  the residual error with  $\epsilon_{itrb} \sim N(0, \sigma_t^2)$  being the residual error for treatment arm t.

In terms of the model parameters the population-level summary for the primary estimand (i.e., the treatment effect at Week 36) can then be expressed as

$$D_{8/3} = \left[\beta_{treat}^{(8mg/3)}\right] - \left[\beta_{treat}^{(2mg)}\right]$$

for the comparison of 8mg/3 with 2 mg and

$$D_{8/5} = \left[\beta_{treat}^{(8mg/5)}\right] - \left[\beta_{treat}^{(2mg)}\right]$$

for the comparison of 8mg/5 with 2 mg.

For this analysis, missing Week 36 BCVA data will be imputed using the Last Observation Carried Forward (LOCF) method. This means that the last non-missing post-baseline BCVA measurement will be carried forward up to Week 36. The summary tables will include the number of participants, least-square mean (LSmean) change (with categorical covariates weighted as observed), unadjusted mean change and standard deviation (SD), as well as the baseline means of each treatment group. For non-inferiority testing, a one-sided alpha of 0.025 will be used for the population-level estimates comparing 2mg Aflibercept Q4 vs (8mg Aflibercept 3xQ4 then Q8) vs (8mg Aflibercept 5xQ4 then Q8).


The results will be presented as LSmean change, the test statistics, degrees of freedom, and corresponding p-values. Additionally, two-sided 95% confidence intervals will be provided. This sensitivity analysis will be performed for the Full Analysis Set (FAS).

# 4.2.3.2 **ANCOVA** with Multiple Imputation

This sensitivity analysis for the primary efficacy endpoint uses ANCOVA after applying multiple imputation to impute missing data (instead of using an LOCF approach). The method follows the same estimand strategy as the primary analysis. The process of multiple imputation involves three steps:

- I. Imputation: Imputation involves generating multiple copies of the original dataset by replacing missing values with appropriate stochastic models. The missing data will be imputed using the Fully Conditional Specification (FCS) method. This method employs an iterative algorithm, where linear regression models are used for prediction and imputation. 10 imputations will be performed using a seed of 22153. The imputation model will include treatment groups, RVO type (CRVO/HRVO vs. BRVO), geographic region (Japan, APAC, Europe, America), categorical baseline BCVA (<60, ≥60), baseline BCVA, and BCVA at each previous post-baseline visit. Imputed values exceeding the normal 0 to 100 range will be truncated to 0 or 100 accordingly.
- II. Analysis: Each of the imputed datasets will be analyzed using ANCOVA, as specified in Section 4.2.3.1. No missing data will be present in the imputed datasets.
- III. Pooling: Pooling combines the different parameter estimates across the imputed datasets based on Rubin's rules (Rubin, 1987) to produce a single point estimate and standard error that takes into account the uncertainty of the imputation process.

This sensitivity analysis will be performed on the Full Analysis Set (FAS).

#### 4.2.3.3 Tipping-point analysis

To evaluate the robustness of the results with regards to departure from the MAR assumption, a tipping-point analysis will be performed based on the results of the multiple imputation analysis described in Section 4.2.3.2. The tipping-point analysis will only be conducted if the multiple imputation analysis demonstrates non-inferiority of the 8 mg groups relative to the 2 mg group.

If non-inferiority can be established, additional tipping-point analyses will be carried out by reducing the imputed BCVA values in the 8mg arms by a series of ascending natural numbers (delta = 1, 2, 3, etc.) with the goal of finding the "tipping point" for each 8mg treatment group that would significantly change the results of the analysis. The smallest delta for which non-inferiority cannot be established will be the "tipping point".

For each delta value, summary tables will include the number of participants, least-square mean change, unadjusted mean change and standard deviation, as well as the baseline means of each treatment group. The estimates will also be expressed as least-square mean change with two-sided confidence intervals at a 5% alpha level, the test statistics, degrees of freedom, and corresponding p-values. This sensitivity analysis will be performed for the FAS.


## 4.2.3.4 Additional Sensitivity Analysis

It has been stated in the CSP Section 9.3.2.3 that an additional sensitivity analysis will be performed to account for important protocol deviations that may potentially affect efficacy for the main analysis of the primary endpoint as described in Section 4.2.2. However, considering the estimand strategy described in Section 1.1, this analysis is deemed obsolete, since relevant ICEs that may potentially affect efficacy are already covered in the estimand definition. Therefore, the sensitivity analysis as described in Section 9.3.2.3 of the CSP will not be performed.

# 4.2.4 Supplementary Analysis

Two supplementary analyses will be conducted based on the supplementary estimands for the primary objective described in Table 1-2.

# **Analysis based on Supplementary Estimand 1:**

A treatment policy strategy will be applied to handle all the ICEs, as presented in Table 1-2, whereby all collected data will be used in the analysis regardless of the occurrence of the ICEs.

For the supplementary estimand, analysis strategies for intercurrent events occurring through Week 36 are described in Table 4-3.

A similar MMRM model as described for the main analysis (Section 4.2.2) will be used to analyze the data. No imputation of missing data will be performed. Missing BCVA measurements will be assumed to be missing at random and will be handled by the MMRM model. No sensitivity analyses will be performed for the supplementary analysis.


Table 4-3: Strategies for occurrence of intercurrent events (ICEs) for analysis at Week 36 for the Supplementary Estimand

| ICE Strategies for the Supplementary Estimand 1 | | |
|---|---|---|
| Intercurrent event | Strategy | Analysis |
| Premature discontinuation of study intervention for any reason before Week 36 | Treatment policy | and discontinuation of study: all observed data will be included in the analysis and the MMRM. Non-observed data beyond discontinuation of study intervention will be assumed to be MAR and will be handled by the MMRM. |
| | | and continuation of study: all observed data will be included in the analysis and the MMRM. |
| Use of a prohibited medication (as defined in section 4.1.7) before Week 36 | Treatment policy | All observed data will be <u>included</u> in the analysis and the MMRM. |
| Missed active injection resulting in an injection interval up to 4 weeks longer than planned | Treatment policy | All observed data will be included in the analysis and the MMRM. |
| Missed active injection resulting in an injection interval more than 4 weeks longer than planned | Treatment policy | All observed data will be <u>included</u> in the analysis and the MMRM. |

# **Analysis based on Supplementary Estimand 2:**

A mixture of treatment policy and composite strategy will be used to handle ICEs, as presented in Table 1-2. Analysis strategies for the occurrence of ICEs are described in Table 4-4.

Table 4-4: Strategies for occurrence of intercurrent events (ICEs) for analysis at Week 36 for the Supplementary Estimand 2

| ICE Strategies for the Supplementary Estimand 2 | | |
|---|---|---|
| Intercurrent event | Strategy | Analysis |
| Premature discontinuation of study intervention due to death before Week 36 | Composite | The change from baseline in BCVA at the visit prior to death will be set to 0. Non-observed data beyond death will be assumed to be MAR and will be handled by the MMRM. |
| Premature discontinuation of<br>study intervention for any other<br>reason than death before Week<br>36 | Treatment policy | and discontinuation of study: all observed data will be included in the analysis and the MMRM. Non-observed data beyond discontinuation of study intervention will be assumed to be MAR and will be handled by the MMRM. and continuation of study: all observed data will be included in the analysis and the MMRM. |
| Use of prohibited medication (as defined in section 4.1.7) before Week 36 | Composite | The change from baseline in BCVA at all visits beyond the first use of prohibited medication through Week 36 will be set to 0. |
| Missed active injection resulting in an injection interval up to 4 weeks longer than planned | Treatment policy | All observed data will be included in the analysis and the MMRM. |
| Missed active injection resulting in an injection interval more than 4 weeks longer than planned | Treatment policy | All observed data will be included in the analysis and the MMRM. |

For participants that experience the intercurrent event "use of prohibited medication" first and discontinue subsequently, the following data rules apply:

- Discontinuation due to death: The change from baseline in BCVA at all visits beyond the first use of prohibited medication through the last visit prior to death will be set to 0 and non-observed data beyond death will not be imputed.
- Discontinuation due to any other reason than death (regardless of whether the participant remained in the study or not): The change from baseline in BCVA at all visits beyond the first use of prohibited medication through Week 36 will be set to 0.

For scenarios where a participant experiences an intercurrent event handled by treatment policy strategy first followed by an intercurrent event handled by composite strategy, the corresponding composite strategy will be applied from the timepoint of the intercurrent event handled by composite strategy as described in the table above.

A similar MMRM model as described for the main analysis (Section 4.2.2) will be used to analyze the data. No imputation of missing data other than the described above will be


performed. Remaining missing BCVA measurements will be assumed to be missing at random and will be handled by the MMRM model. No sensitivity analyses will be performed for the supplementary analysis.

#### 4.3 Secondary Endpoints Analysis

## 4.3.1 Key Secondary Endpoint

## **4.3.1.1 Definition of Endpoint(s)**

The key secondary efficacy endpoint in this study is the number of active injections from baseline to Week 64. Active injections refer to the number of injections that were actually administered, as opposed to the number of planned injections.

In addition to the number of injections that were actually administered, the endpoint value will also reflect the occurrence of certain intercurrent events: premature discontinuation of study intervention due to a treatment-related adverse event or lack of efficacy, which will be addressed using a composite and a hypothetical strategy, respectively. Participants experiencing these types of intercurrent events will have their endpoint value calculated in a way that reflects an unfavorable outcome (under the composite strategy) or an injection schedule under a hypothetical scenario. See Section 4.3.1.3 for details.

### 4.3.1.2 Main Analytical Approach

The analysis will be conducted in a pairwise manner, i.e., comparing the 8 mg/3 treatment group vs the 2 mg treatment group and the 8 mg/5 treatment group vs the 2 mg treatment group in two separate analyses. For simplicity, in the following the secondary analysis will be formulated in a general manner and applied to both pairwise comparisons of 8 mg/3 treatment group vs the 2 mg treatment group and 8 mg/5 treatment group vs the 2 mg treatment group.

The key secondary endpoint, the number of active injections from baseline to Week 64, will be analyzed using a non-parametric rank analysis of covariance (non-parametric rank ANCOVA). This analysis will adjust for covariates when comparing treatment groups. Additionally, treatment effects will be estimated using a linear regression model adjusted for the same covariates.

Endpoint values will be unobservable (missing) for participants who prematurely discontinue the study intervention due to reasons other than treatment-related adverse events or lack of efficacy. Their treatment schedule will be modeled under a hypothetical scenario as discussed in Section 4.3.1.3. No other type of missing data is expected for this endpoint.

To impute hypothetical values, a MI model (Rubin, 1987) will be employed. The process involves creating multiple imputed datasets, and each dataset will be subjected to the same analysis procedures using the non-parametric rank ANCOVA and linear regression. The results from multiple imputed datasets will then be combined for overall inference using the Rubin's rule. Each of the steps mentioned above is described in more detail below.

Missing endpoint values (total number of active injections) for participants with aforementioned intercurrent events will be imputed in alignment with the hypothetical scenario, namely that these participants would receive a similar number of active injections as other participants without such intercurrent events with similar baseline characteristics within their treatment arm. The imputation model will include as predictors the same baseline covariates as those included in the analysis models described below, i.e., baseline BCVA, baseline CST, and the stratification factors for region, BCVA score (greater equal than or less than 60), and


RVO type. The stratification variable 'region' will be collapsed into three categories (Japan+APAC, Europe, and America) by combining the two smaller strata Japan and APAC. This adjustment is made because the rank ANCOVA is a randomization-based method with variance estimation under the null hypothesis of no treatment difference in all strata. The asymptotic statistical properties of this approach rely on the central limit theory, which conventionally requires approximately 30 samples in each stratum (Gasparyan, 2021) to support its statistical properties. The Predictive Mean Matching imputation method (Heitjan and Little 1991; Schenker and Taylor 1996) will be used, which will ensure that the imputed values are integer and in the range of allowed number of injections within each treatment arm. The number of donor observations, a user-specified parameter of the Predictive Mean Matching imputation method, will be set to 5 (default in SAS Proc MI).

To ensure robustness, a total of 500 multiple imputation steps will be conducted.

The MI model will be implemented as follows, using the SAS pseudo code given below as an example. Alternatively, R may be used for the actual analysis. The random seed (22153) will be specified in the corresponding option of Proc MI in SAS or its equivalent in R.

```
/* Step 1: Perform multiple imputation */
proc mi data=my_data out=multiple_imputed_data seed=22153 nimpute=500;
  class treatment region_RVO_BCVA;
  var baseline_BCVA baseline_CST treatment region_RVO_BCVA active_injections;
  monotone regpmm (active_injections / k=5);
run;
```

where "region\_RVO\_BCVA" is a categorical variable with 12 levels, representing a cross of the three original stratification factors baseline BCVA score, region (collapsed into three categories as described above), and RVO type.

For the non-parametric ANCOVA, the Cochran-Mantel-Haenszel score test will be applied to residuals of a regression model on rank-transformed data as described in <u>Stokes et al. (2012)</u>. Baseline BCVA, baseline CST, and the stratification factors region (collapsed to three categories as describe above), BCVA score (greater equal than or less than 60), and RVO type will be adjusted for.

The methodology described by <u>Stokes et al. (2012)</u> will be applied as follows (and exemplified based on the SAS pseudo code provided below). First, the endpoint values (total number of injections) and continuous baseline covariates baseline BCVA and baseline CST will be transformed to standardized ranks by stratum using fractional ranks and the mean method for ties will be implemented as:

Subsequently, separate regression models will be fit within each stratum defined by the stratification factors, using the standardized rank values of the endpoint as dependent and of


the baseline BCVA and CST values as independent variables, respectively. Residuals from these models will be captured for further testing of differences between treatment groups:

Finally, the stratified Cochran-Mantel-Haenszel (CMH) mean score test, using the residuals as scores, will be used to compare the two treatment groups as:

```
/* Step 4: Implement the Cochran-Mantel-Haenszel (CMH) test */
proc freq data=residuals;
  by _Imputation_;
  tables region*BCVA_score*RVO_type*treatment*resid / CMH2;
  ods output cmh=cmhstat;
run:
```

The non-parametric rank ANCOVA described above will be applied to each imputation dataset within the multiple imputation procedure. Before combining the results of the CMH test using Rubin's rule, a normalizing transformation using the Wilson-Hilferty transformation, as described in Ratitch et al. (2013), will be applied. The CMH statistic computed for each imputed dataset ( $cmh^{(m)}$ ) will be standardized using its corresponding degrees of freedom (df) to obtain the standardized test statistic  $st\_cmh^{(m)}$  as:

$$st\_cmh^{(m)} = \frac{\sqrt[3]{\frac{cmh^{(m)}}{df}} - \left(1 - \frac{2}{9 \times df}\right)}{\sqrt{\frac{2}{9 \times df}}}$$

```
/* Step 5: Standardize the CMH statistic for each imputed dataset */
data cmh_stat;
  set cmhstat;
  std_cmh = ((cmh/df)**(1/3) - (1-2/(9*df))) / sqrt(2/(9*df));
  std_cmh_stderr = 1;
run;
```

The standardized statistic, along with its standard error of 1, will be used to perform a combined CMH test using Rubin's rule as:

```
/* Step 6: Perform the combined CMH test using Rubin's rule */
proc mianalyze data=cmh_stat;
  modeleffects std_cmh;
```


Along with evaluating the treatment effect based on the non-parametric rank ANCOVA for each pairwise comparison (i.e., 8mg/3 vs 2mg and 8mg/5 vs 2mg), a single linear regression model including the treatment group variable with three levels (2mg vs 8mg/3 vs 8mg/5) and adjusted for baseline BCVA, baseline CST, and the stratification factors region (collapsed to three categories Japan+APAC, Europe, and America as described above), BCVA score (greater equal than or less than 60), and RVO type will be used to estimate the treatment effects. The linear regression model can be represented by the following formula:

$$y = \beta_0 + \beta_1 x_1 + \beta_2 x_2 + \beta_3 x_3 + \beta_4 x_4 + \beta_5 x_5 + \beta_6 x_6 + \varepsilon \quad (1)$$

Where:

- y is the response variable (i.e. number of active injections from baseline to Week 64),
- $\beta_0$  is the intercept,
- $x_1, x_2$ , and  $x_3$  are the region, BCVA score, and RVO type variables.
- $x_4$ , and  $x_5$  are the baseline variables (Baseline BCVA and Baseline CST)
- $x_6$  is the treatment group variable (i.e. 2mg vs 8mg/3 vs 8mg/5),
- $\beta_1, \beta_2, \beta_3, \beta_4$  and  $\beta_5$  are the corresponding regression coefficients for the stratification factors and baseline variables,
- $\beta_6$  represents the regression coefficient for the treatment group variable, and
- $\varepsilon$  is the error term.

In terms of the model parameters the population-level summary for the secondary estimand (i.e., the number of injections at week 64) can then be expressed as

$$D_{8/3} = \left[\beta_{6}^{(8mg/3)}_{treat}\right] - \left[\beta_{6}^{(2mg)}_{treat}\right]$$

for the comparison of 8mg/3 with 2 mg and

$$D_{8/5} = \left[\beta_{treat}^{(8mg/5)}\right] - \left[\beta_{6treat}^{(2mg)}\right]$$

for the comparison of 8mg/5 with 2 mg.

Please note that this formulation is intended as a general framework. For each categorical variable (Region, BCVA score, and RVO type), the model will include p-1 coefficient estimates, where p corresponds to the number of categories within the variable. Furthermore, a separate variance term will be estimated for each treatment group. The linear regression model will be fit to each of the imputation data sets created in the previous step. The treatment effect estimate across the imputation datasets will be then combined using Rubin's rule and the corresponding 95% confidence interval will also be created.

For cases where the baseline CST measurement is not available from the reading center, the investigator assessment of the baseline CST will be used in the analysis of the number of active injections described in this section.


The two-sided p-value based on the non-parametric rank ANCOVA, as well as the linear regression treatment estimates (with categorical covariates weighted as observed) together with the corresponding standard error and 95 % confidence interval, will be reported.

Descriptive summary tables will be provided by treatment group for:

• All observed cases regardless of the occurrence of an ICE in the FAS population

#### 4.3.1.3 Strategies for occurrence of intercurrent events

Analysis strategies for intercurrent events for the secondary estimand occurring before week 64 are described in Table 4-6 below.

For the intercurrent event "Premature discontinuation of study intervention due to lack of efficacy", a hypothetical strategy will be applied assuming that the patient would have continued in the study and would have met the DRM criteria for shortening at each active injection visit. The number of injections administered until the occurrence of the intercurrent event will be counted. After the occurrence, it will be assumed that the patients would have continued to be treated as often as possible according to the DRM criteria, i.e., meeting the shortening criteria at every visit with an active injection after the occurrence of the ICE. For example, as shown in Table 4-5, if a participant discontinues due to LoE while on an 8-week interval, for example, his/her next injection would be as scheduled, but then the interval will be shortened to 4 weeks, and the participant will be treated every 4 weeks thereafter. Specifically, as shown in Table 4-5, if Patient 1 discontinues due to LoE at week 20, it will be assumed that his/her following dosing intervals will be shortened to 4 weeks, thus receiving additional active doses at Week 28 and remaining on 4-week intervals until the end of the study. Similarly, if Patient 2 discontinues due to LoE while on a 12-week interval at week 44, it will be assumed that his/her following dosing interval will be shortened to 8 weeks, thus receiving additional active doses at Week 52 and then shortened again to 4-week intervals and subsequently remaining on 4-week intervals until the end of the study.

**Table 4-5: Shortening Criteria** 



This approach would ensure that none of the affected participants can have missing data and reflects what could have happened if the participant had remained in the study.


Table 4-6: Strategies for occurrence of intercurrent events for analysis at week 64 for the Secondary Estimand

| ICE Strategies for Secondary Estimand | | |
|---|---|---|
| Intercurrent event | Strategy | Secondary Analysis |
| Premature discontinuation of study intervention due to lack-of-efficacy | Hypothetical | See details in text above. |
| Premature discontinuation of study intervention due to treatment related AEs | Composite | Discontinuations due to treatment related AE is considered as treatment-failure and the number of injections will be set to 16 to represent an unfavorable outcome |
| Premature discontinuation of study intervention due to treatment unrelated AEs and other reasons | Hypothetical | Non-observed data beyond discontinuation of study intervention due to treatment unrelated AEs and other reasons will be imputed using multiple imputation technique as described in Section 4.3.1.2. |
| Missed injection | Treatment policy | The observed number of injections will be used in the analysis. |

### 4.3.1.4 Supplementary Analyses

The analysis presented in Section 4.3.1.2 will be repeated for the subgroup of participants who completed the study intervention period, that is, for the participants that did not prematurely discontinue study intervention (for any reason) prior to the end of study at week 64. In this particular subgroup, the intercurrent event strategies for premature discontinuation of study intervention as outlined in Table 4-6 will not be applicable. Moreover, complete data on the number of injections at Week 64 will be accessible for all participants. Consequently, there won't be any missing data issues related to the number of injections, and the multiple imputation method detailed in Section 4.3.1.2 will not be used.

The nonparametric rank ANCOVA and the linear regression model for estimating the treatment effect, as described in Section 4.3.1.2, will be applied to this subgroup. A 95% CI based on the linear regression model will be provided along with a 95 % CI based on bootstrapping. The bootstrap confidence interval will be constructed generating B=1000 bootstrap samples by fitting the linear regression model to each bootstrap sample and obtaining B treatment effect estimates. The final bootstrap confidence interval will be constructed using the basic percentile method where the 2.5th and 97.5th percentiles of the B treatment effect estimates defining the limits of the confidence interval (Efron and Tibshirani 1993). Bootstrap samples will be drawn with replacement from the observed data of the subgroup.

#### 4.3.2 Supportive Secondary Endpoints

The following additional secondary efficacy endpoints will be evaluated:


- Number of active injections from baseline to Week 36
- Change from baseline in BCVA measured by the ETDRS letter score at Week 44 for the 8mg/5 and 2 mg groups only.
- Change from baseline in BCVA measured by the ETDRS letter score at Week 64.
- Participant gaining at least 15 letters in BCVA from baseline at Weeks 36 and 64.
- Participant achieving an ETDRS letter score of at least 69 (approximate 20/40 Snellen equivalent) at Weeks 36 and 64.
- Participant having no IRF and no SRF in the center subfield at Weeks 36 and 64.
- Change from baseline in CST at Weeks 36 and 64.
- Change from baseline in NEI-VFQ-25 total score at Weeks 36 and 64.
- Participants dosed only Q8W through Week 36 in the 8 mg Q8W group.
- Participant having last treatment interval ≥12 or of 16 weeks at Week 64.
- Participant having next intended interval  $\ge 12, \ge 16$  or of 20 weeks at Week 64.

All analyses will be conducted on the FAS. Unless specified otherwise, summary statistics (see also Section 4.1) will be provided by treatment group and visit for:

- for all observed cases regardless of the occurrence of an ICE
- for all observed cases until the occurrence of an ICE in line with the primary estimand strategy.

Unless otherwise stated, the main evaluation of the binary secondary endpoints will be based on the summary statistics in line with the primary estimand strategy.

### 4.3.2.1 Number of active injections from baseline to Week 36

The number of active injections from baseline to Week 36 will be analyzed descriptively by treatment group and by using the analysis described for the key-secondary endpoint in Section 4.3.1. Intercurrent events will be handled similarly as described in Table 4-6. However, for the composite strategy for the ICE "premature discontinuation of study intervention due to treatment related AEs" the value for the number of injections will be set to 9 (the maximum possibly by Week 36). This analysis will be performed once all participants have completed Week 36 or have discontinued the study prematurely. Summary statistics will be presented by treatment group in line with the key-secondary endpoint described in Section 4.3.1.2.

## 4.3.2.2 Change from baseline in BCVA measured by the ETDRS letter score at Week 44 for the 8mg/5 and 2 mg groups only

The endpoint of "Change from baseline in BCVA measured by the ETDRS letter score at Week 44 for the 8mg/5 and 2 mg groups only" will be analyzed descriptively by treatment group and using the mixed model for repeated measurements (MMRM) as described in Section 4.2.2. The MMRM analysis will include baseline BCVA measurement as a covariate and treatment group, visit, and stratification variables (geographic region, categorized baseline BCVA, and RVO type) as fixed factors. Additionally, terms for the interaction between baseline and visit and for the interaction between treatment (8mg/5 and 2 mg groups only) and visit (up to week 44) will also be included in the analysis.


## 4.3.2.3 Change from baseline in BCVA measured by the ETDRS letter score at Week 64.

The endpoint of "Change from baseline in BCVA measured by the ETDRS letter score at Week 64" will be analyzed descriptively by treatment group and using the mixed model for repeated measurements (MMRM) as described in Section 4.2.2. The MMRM analysis will include baseline BCVA measurement as a covariate and treatment group, visit, and stratification variables (geographic region, categorized baseline BCVA, and RVO type) as fixed factors. Additionally, terms for the interaction between baseline and visit and for the interaction between treatment and visit (up to week 64) will also be included in the analysis.

## 4.3.2.4 Participant gaining at least 15 letters in BCVA from baseline at Weeks 36 and 64.

The proportion of participant gaining at least 15 letters in BCVA from baseline at Weeks 36 and 64 will be analyzed descriptively. Missing cases will not be included in the denominator when calculating proportions.

# 4.3.2.5 Participant achieving an ETDRS letter score of at least 69 (approximate 20/40 Snellen equivalent) at Weeks 36 and 64.

The proportion of participants achieving an ETDRS letter score of at least 69 at Week 36 and 64 will be analyzed descriptively. Missing cases will not be included in the denominator when calculating proportions.

## 4.3.2.6 Participant having no IRF and no SRF in the center subfield at Weeks 36 and 64.

The proportion of participants having no IRF and no SRF in the center subfield at Weeks 36 and 64 will be analyzed descriptively. Missing cases will not be included in the denominator when calculating proportions.

#### 4.3.2.7 Change from baseline in CST at Weeks 36 and 64.

The endpoints "Change from baseline in CST measured at Week 36" and "Change from baseline in CST measured at Week 64" will be analyzed both descriptively by treatment group and using the mixed model for repeated measurements (MMRM) as described in Section 4.2.2. The MMRM analysis will include baseline CST measurement as a covariate and visit, treatment group and stratification variables (geographic region, categorized baseline BCVA, and RVO type) as fixed factors. Additionally, terms for the interaction between baseline and visit and for the interaction between treatment and visit (up to Week 36 and Week 64) will also be included in the analysis.

## 4.3.2.8 Change from baseline in NEI-VFQ-25 total score at Weeks 36 and 64.

The change from baseline in NEI-VFQ-25 total score at Weeks 36 and 64 will be analyzed both descriptively by treatment group and using the ANCOVA using LOCF approach as described in Section 4.2.3.1 based on the sensitivity analysis strategy for the primary estimand. The ANCOVA analysis will include baseline NEI-VFQ-25 total score measurement as a covariate and treatment group, visit, and stratification variables (geographic region, categorized baseline BCVA, and RVO type) as fixed factors.


## 4.3.2.9 Participants dosed only Q8W through Week 36 in the 8 mg Q8W group.

The number participants dosed only Q8W through Week 36 in the 8 mg Q8W group will be provided as part of the exposure analysis as described in Section 6.1.3.

## 4.3.2.10 Participant having last treatment interval ≥12 or of 16 weeks at Week 64.

The proportion of participants having last treatment interval  $\geq$ 12 or of 16 weeks at Week 64 will be provided as part of the exposure analysis as described in Section 6.1.3.

## 4.3.2.11 Participant having next intended interval ≥12, ≥16 or of 20 weeks at Week 64.

The proportion of participants having next intended interval  $\ge 12$ ,  $\ge 16$  or of 20 weeks at Week 64 will be provided as part of the exposure analysis as described in Section 6.1.3.

#### 4.3.2.12 Pharmacokinetics

**Endpoint:** Systemic exposure to aflibercept as assessed by plasma concentrations of free, adjusted bound and total aflibercept from baseline through Weeks 36 and 64.

All the analyses performed for PK samples will be carried out by treatment group on the PKS analysis set. This study does not evaluate any pharmacodynamic parameters.

PK samples are collected at baseline (Visit 2), Week 4 (Visit 3), Week 12 (Visit 5), Week 16 (Visit 6), Week 24 (Visit 8), Week 36 (Visit 11) and Week 64 (Visit 18) for all participants. The individual concentrations of free, adjusted bound, and total aflibercept over time will be summarized and listed by descriptive statistics by visit.

Individual concentrations of adjusted bound aflibercept will be calculated as 0.717 x individual concentrations of bound aflibercept.

Individual concentrations of total aflibercept will be calculated as the sum of individual concentrations of free and adjusted bound aflibercept.

The following LLOQs are used by the laboratory:

- For free aflibercept assay: LLOQ = 15.6ng/mL
- For bound aflibercept assay: LLOQ = 31.3ng/mL

Drug concentrations will be further grouped by the following baseline factors:

- age categories as defined in Section 6.1.1,
- medical history of renal impairment as determined by baseline serum creatinine values as defined in Section 6.3.6,
- hepatic impairment based on medical history as defined in Section 6.3.7,
- BMI categories as defined in Section 6.1.1,
- ethnicity as defined in Section 6.1.1,
- race grouped as White, Asian, Black or African American, and Other/Not Reported,

and evaluated by means of descriptive statistics.

No formal statistical hypothesis testing will be performed.


### 4.4 Exploratory Endpoints Analysis

The following exploratory endpoints will be analyzed using descriptive statistical methods by treatment group.

Unless specified otherwise, summary statistics (see also Section 4.1) will be provided by treatment group and visit for:

- for all observed cases regardless of the occurrence of an ICE
- for all observed cases until the occurrence of an ICE in line with the primary estimand strategy.

The exploratory endpoints are:

## 4.4.1 Change from baseline in BCVA measured by the ETDRS letter score at each visit

The exploratory endpoint of "Change from baseline in BCVA measured by the ETDRS letter score at each visit" will be analyzed descriptively by treatment group.

## 4.4.2 Participant with vision changes of at least 5, 10, or 15 letters in BCVA from baseline at each visit

The proportion of participants with vision changes of at least 5, 10, or 15 letters in BCVA from baseline at each visit will be analyzed descriptively. Missing cases will not be included in the denominator when calculating proportions.

#### 4.4.3 Participant with no IRF and no SRF in the center subfield at each visit

The proportion of participants with no IRF and no SRF in the center subfield at each visit will be analyzed descriptively. Missing cases will not be included in the denominator when calculating proportions.

## 4.4.4 Time to fluid-free retina over 36 and 64 weeks (total fluid, IRF, and/or SRF in the center subfield)

Total fluid-free retina (no IRF and no SRF in central subfield) is defined as the absence of total fluid, i.e. no IRF and no SRF in the central subfield as found in the SD-OCT, regardless of whether any retinal fluid was found again after that.

Time to total fluid-free retina (no IRF and no SRF in central subfield) will be analyzed by Kaplan-Meier analysis and shown in Kaplan-Meier plots and descriptive summaries. Estimated event rates at Week 36 and Week 64 will be provided along with the Hazard Ratios (HRs) and p-values. Time to total fluid-free retina is defined as the duration from randomization to the timepoint when total fluid was absent for the first time whereas intercurrent events are handled according to Table 6-11. The analysis will be performed using the study visits (i.e. multiples of 4 weeks) and not the calendar time as unit. Participants without total fluid-free retina will be censored at the time of their last SD-OCT assessment.

HRs will be calculated using a stratified Cox proportional hazards model, including treatment group as a factor and stratification variables. The p-value will be calculated by a stratified log-rank test to compare the 8mg groups vs. the 2mg group.


Time to IRF-free retina (no IRF in central subfield) and time to SRF-free retina (no SRF in central subfield) will be analyzed in the similar way.

Participants with no fluid at baseline are considered to not be "at risk" and are thus excluded from the analysis. Similarly, participants with missing baseline information or with baseline category "undetermined" for the fluid status (see Section 4.1.6) are also excluded. If both IRF status and SRF status are undetermined, then the total fluid-free retina status is also undetermined.

## 4.4.5 Participant having sustained fluid-free retina over 36 and 64 weeks (total fluid, IRF, and/or SRF in the center subfield)

Sustained total fluid-free retina (no IRF and no SRF in central subfield) is defined as the absence of total fluid for at least 2 consecutive visits and all subsequent visits, i.e. no IRF and no SRF in the central subfield as found in the SD-OCT. The proportion participants having sustained fluid-free retina over 36 and 64 weeks (total fluid, IRF, and/or SRF in the center subfield) will be analyzed descriptively. Missing cases will not be included in the denominator when calculating proportions.

### 4.4.6 Change in area of retinal ischemia at Weeks 36 and 64

The change in area of retinal ischemia at Weeks 36 and 64 will be analyzed descriptively by treatment group.

## 4.4.7 Change in the area of fluorescein leakage at Weeks 36 and 64.

The change in the area of fluorescein leakage at Weeks 36 and 64 will be analyzed descriptively by treatment group.

#### 4.5 Safety Analyses

The analysis of safety variables will be performed descriptively on the SAF population at Weeks 36 and 64. The data collected at these timepoints will be used to generate descriptive statistics as described in Section 4.1 for continuous and categorical data. The purpose of this analysis is to provide an overview of the safety data, including the occurrence of adverse events, serious adverse events, and other safety-related variables. This may involve transforming the data or utilizing categorical cut-points for safety scales to enhance our understanding of safety trends.

#### 4.5.1 Adverse Events

The analysis of adverse events (AEs) will be conducted according to the following procedures:

- An AE is defined as any adverse medical event in a study participant that is associated with the use of study intervention, regardless of its relation to the study intervention.
- All reported AEs will be coded using the latest version of MedDRA at the time of database lock. Coding will be done at the lowest level of specificity according to Bayer's global standards.
- AEs will be recorded from the time of informed consent signature until the end of the study. If a participant withdraws from the study during the screening process, AEs will


be recorded up until their withdrawal. If a participant is withdrawn after receiving the first dose of study medication, AEs will be recorded up until 30 days after their last dose of study intervention or the termination visit, whichever is later.

• A Treatment-emergent adverse events (TEAE) are defined as AEs that occurred in the time frame from first injection (active or sham) to the last injection (active or sham) plus 30 days. For the participants who have not discontinued study treatment prematurely (i.e., are "ongoing") at the Week 36 analysis, all AEs that started at first injection or later will be considered treatment-emergent.

The data cut-off rules for Week 36 and Week 64 AE reporting are described in a separate document ("Data Cut-Off Specifications").

The proportions of participants experiencing AEs will be used as safety variables for AE summary. Other variables used for AE description and analysis will include AE Verbatim Term, AE start date/time and end date/time/ongoing, corresponding study day, AE Duration, relationship of AE to study drug, relationship of AE to commercial aflibercept (2 mg), relationship of AE to intravitreal injection, relationship of AE to protocol-required procedure, seriousness, intensity, action due to AE, treatment of AE, and outcome. Summaries that include frequencies and proportions of participants reporting AEs will include the Preferred Terms (PTs) and the System Organ Classes (SOCs).

Evaluations for TEAEs will mainly be conducted for the following categories, which will be identified from the information in the Case Report Form (CRF):

- Ocular TEAEs in the treated study eye
- Ocular TEAEs in the fellow eye
- Non-ocular TEAEs

AE summaries will be provided, displaying AEs within each SOC in alphabetical order. For an overall characterization of the AE profile for aflibercept in this study, an AE summary will include AEs within each SOC listed in alphabetical order, with columns for treatment groups, including a column "All 8mg" for the pooled 8mg group.

TEAEs in the study eye assessed by the investigator as being related to the injection procedure, related to protocol-required procedures, and those related to the study medication will be summarized separately. TEAEs in the fellow eye assessed by the investigator as being related to the injection procedure, related to protocol-required procedures, related to the study medication, and those related to commercial aflibercept (2 mg) will also be summarized separately.

A listing will be constructed that includes the participant identification, treatment group, category of AE (ocular study eye, non-ocular), AE, MedDRA term, seriousness, severity, causality, elapsed time to onset since first dose of aflibercept and since last does of aflibercept, duration, and outcome.

**Serious Adverse Events (SAEs)** will be summarized in the same way as described for TEAEs.

A frequency table of TEAEs of intraocular inflammation of study eye terms, crosstabulated with related MedDRA PT and SOC, will be displayed by treatment arm (see Section 6.3.2 for the definition of terms).


A frequency table of adjudicated treatment-emergent Anti-Platelet Trialists Collaboration (APTC) events terms, cross-tabulated with related MedDRA PT and SOC, will also be displayed by treatment arms. The adjudication of AE is described in the "APTC adjudication committee charter".

Additionally, frequency tables of TEAEs of **hypertension** terms and **nasal mucosal finding** terms, cross-tabulated with related MedDRA PT and SOC, will be displayed by treatment arm (see Section 6.3 for the definition of terms).

Adverse Event of Special Interest (AESI) as defined in the study protocol are arterial thromboembolic events including cerebrovascular ischemic events and cardiovascular ischemic events and will be summarized in the same way as described for TEAEs.

#### 4.5.1.1 Subgroup Analyses

Subgroup analyses for TEAEs will be performed for the safety analysis subgroups described in Section 4.6.1 and by RVO type as describe in Section 4.6.2 for each of the following types of TEAE:

Number of participants with

- ocular TEAEs in the study eye
- non-ocular TEAEs
- Serious ocular TEAEs in the study eye
- Serious non-ocular TEAEs

#### 4.5.2 Additional Safety Assessments

#### 4.5.2.1 Surgeries

All surgeries after informed consent will be collected on the CRF, and a listing of all surgeries and diagnostic procedures will be provided.

#### 4.5.2.2 Clinical Laboratory Variables

Chemistry, hematology, and urinalysis will be collected at screening (Visit 1), Week 36 (Visit 11), and Week 64 (EOS) or ED. Pregnancy testing will be performed at each visit. The tests detailed in Table 4-7 will be conducted by the central laboratory.


Table 4-7: Pre-defined laboratory abnormalities

| Laboratory | Parameters | |
|---|---|---|
| <b>Assessments</b> | | |
| Hematology | Platelet count | WBC count |
| | RBC count | Differential: |
| | Hemoglobin | Neutrophils |
| | Hematocrit | Lymphocytes |
| | RBC Indices | Monocytes |
| | | Eosinophils |
| | | Basophils |
| Clinical Chemistry | | Total and direct bilirubin |
| | Potassium | Urea (or BUN) |
| | Chloride | LDH |
| | Carbon dioxide | Total protein, serum |
| | Calcium | Total cholesterol |
| | Creatinine | Triglycerides |
| | Glucose (non-fasting) | LDL |
| | Albumin | HDL |
| | AST/SGOT | Uric acid |
| | ALT/SGPT | CPK |
| D. C. Historia | Alkaline phosphatase | |
| Routine Urinalysis | 1 0 1, 1 | |
| | | ), protein, blood, ketones, bilirubin, nitrite, |
| | leukocyte esterase by di | • |
| | | other casts, bacteria, epithelial cells, yeast |
| | <ul> <li>Creatinine</li> </ul> | |
| | <ul><li>UPCR</li></ul> | |
| Other Screening | <ul> <li>Follicle stimulating hormone and estradiol (as needed in women of non-<br/>childbearing potential only)</li> </ul> | |
| Tests | | |
| | <ul> <li>Highly sensitive serum h</li> </ul> | CG pregnancy test (as needed for WOCBP) <sup>a</sup> |

ALT=alanine aminotransferase, AST=aspartate aminotransferase, BUN=blood urea nitrogen, CPK=creatine phosphokinase, eCRF=electronic Case Report Form, hCG=human chorionic gonadotropin, HDL=high density lipoprotein, LDH=lactate dehydrogenase, LDL=low density lipoprotein, RBC=red blood cell, SGOT=serum glutamic-oxaloacetic transaminase, SGPT=serum glutamic-pyruvic transaminase, UPCR=urine protein: creatinine ratio, WBC=white blood cell, WOCBP=women of childbearing potential

For WOCBP, a negative serum pregnancy test at screening is required for eligibility.

Number and percentage of participants with a treatment-emergent potentially clinically significant value (PCSV, any value fulfilling pre-defined criteria for abnormal laboratory parameters as described in Table 6-1 in the Appendix 6.2) at any time point will be summarized for selected clinical laboratory test for all participants.

Laboratory values out of normal range will be summarized in tables and also flagged in laboratory value listings.

#### 4.5.2.3 Electrocardiogram

A standard digital 12-lead Electrocardiogram (ECG) will be performed at screening (Visit 1), Week 36 (Visit 11), and Week 64 (EOS) or ED. ECG variables, including heart rate, PR interval, QRS duration, RR interval, QT interval, and overall interpretation of ECG (normal/abnormal), will be analyzed for the SAF using appropriate descriptive methods.


Change from baseline or frequency tables and/or cross-tabulation of baseline vs. post-baseline status for categorical variables (overall interpretation of ECG normal/abnormal) will be presented by visit and treatment arms. QTc with Bazett and Fridericia correction will be used.

### 4.5.2.4 Vital Signs

Vital signs, including heart rate, systolic blood pressure, and diastolic blood pressure, will be collected pre-injection and before any blood draws at each visit during the study. The timing of blood pressure assessments should be within ±2 hours of the clock time of dosing at the baseline visit, if possible. Vital signs will be summarized by baseline and change from baseline to each scheduled visit by treatment group for the SAF.

Additionally, summaries will be provided for participants with at least one treatmentemergent PCSV of systolic blood pressure:

- $\leq$  95 mmHg and decrease from baseline  $\geq$  20 mmHg
- $\geq$ 160 mmHg and increase from baseline  $\geq$  20 mmHg

As well as for participants with diastolic blood pressure treatment emergent PCSV of

- $\leq$  45 mmHg and decrease from baseline  $\geq$  10 mmHg
- $\geq$ 110 mmHg and increase from baseline  $\geq$  10 mmHg.

Heart rate and blood pressure assessments will also be displayed as figures with mean change from baseline for SAF.

## 4.5.2.5 Other Safety Measures

Variables of analysis for ocular safety measures include:

- Proportion of participants with increased IOP
  - $\circ$   $\geq$  10 mmHg increase in IOP measurement from baseline to any pre-dose measurement
  - > 21 mmHg for any pre-dose measurement at any time during the study
  - $\circ$   $\geq$  25 mmHg for any pre-dose measurement at any time during the study
  - $\circ \geq 35$  mmHg for any pre-dose or post-dose measurement at any time during the study,

where the post-dose IOP measurement will be the final measurement before the participant leaves the site.

Summary statistics will also be displayed by visit for:

- change from baseline for pre-dose IOP values
- Proportion of participants with Anterior Chamber Cells (only pre-dose assessment for study eye)
  - o 0: no cells
  - o Trace: less than 5 cells
  - o 1+: 5 to 10 cells
  - o 2+: 10 to 20 cells


- o 3+: 20 to 30 cells
- o 4+: cells too numerous to count.
- Proportion of participants with Anterior Chamber Flare (only pre-dose assessment for study eye)
  - o 0: no protein
  - Trace: trace amount of protein
  - o 1+: mild amount of protein
  - o 2+ and 3+: moderate amount of protein (continuum)
  - o 4+: severe amount of protein.

Frequency tables will be provided for each of the above categories at each visit where data is available. Shift tables will be provided for the gradings (only pre-dose assessment for study eye).

- Portion of participants with retinal ischemia (perifoveal and parafoveal ischemia, non-perfusion outside the macula) by FA
- Portion of participants with macular leakage by FA

Frequency tables will be provided for each of the above categories at each visit where data is available.

#### 4.6 Other Analyses

#### 4.6.1 Subgroup Analyses

Exploratory subgroup analyses will be performed, using descriptive summary statistics for the following subgroups:

- 1. Age at enrollment: < 55 years,  $\ge 55$  to < 65 years,  $\ge 65$  years to < 75 years,  $\ge 75$  years
- 2. Sex: male, female
- 3. Geographic region:
  - Japan vs. APAC vs Europe vs America
  - USA vs Rest of the world
  - Asia (Japan and APAC) vs ROW
- 4. Ethnicity: Not Hispanic or Latino, Hispanic or Latino
- 5. Race (only categories with sufficient sample size): Asian, White
- 6. Baseline BCVA: < 60 letters,  $\ge 60$  letters
- 7. Baseline CST:  $\leq$  observed median, > observed median
- 8. Medical history of hypertension: No, Yes (see section 6.3.1)
- 9. Medical history of diabetes: No, Yes
- 10. Medical history of cerebrovascular disease: No, Yes (see section 6.3.4)
- 11. Medical history of ischaemic heart disease: No, Yes (see section 6.3.5)


- 12. Medical history of renal impairment: Normal, Mild, Moderate, Severe (see section 6.3.6)
- 13. Medical history of hepatic impairment: No, Yes (see section 6.3.7)

Subgroups 1 to 7 will be analyzed for the primary and key secondary endpoints. For subgroup analysis based on geographic regions and categorized baseline BCVA, the corresponding variable will be excluded from the statistical models. These subgroup analyses are exclusively descriptive, and tables will present 95% confidence intervals. For the primary endpoint, subgroups will be analyzed using the MMRM without imputing missing values (see Section 4.2.2), for the key-secondary endpoint, subgroups will be analyzed using the non-parametric rank ANCOVA (see Section 4.3.1.2). In the subgroup analyses of the key-secondary endpoint, the stratification factor "region" will be excluded from the analysis and imputation model to mitigate issues associated with small sample sizes within strata. Subgroups 1 to 13 will be analyzed for the safety analyses mentioned in Section 4.5.1.1.

If the number of participants in a subgroup is less than 10%, the subgroup categories may be redefined prior to unmasking.

### 4.6.2 Subgroup Analysis by RVO type

To conduct a supportive exploratory subgroup analysis for BRVO and CRVO/HRVO, we plan to randomize a minimum of 40% of participants (i.e., 329 participants) per RVO type ([CRVO or HRVO] vs BRVO).

The primary efficacy endpoint will be analyzed for the FAS, as described in Section 4.2.2, by RVO type (CRVO/HRVO or BRVO) and by:

- individual arm (2q4 vs 8q8/3 vs 8q8/5)
- pooling the two 8mg arms (8q8/3 and 8q8/5).

The corresponding RVO type variable will be excluded from the MRMM statistical model, and for the analysis with pooled 8mg arms the treatment group variable will only consist of two categories (8mg vs 2mg).

Furthermore, summary statistics for the subgroup analysis by RVO type (CRVO/HRVO or BRVO) will be presented.

Furthermore, the secondary endpoint "Number of active injections from baseline to Week 36" will also by analyzed as described in Section 4.3.2.1 by RVO type (individual arms). For the secondary endpoints "Change from baseline in CST at Weeks 36 and 64", descriptive summary statistics by RVO type will be provided.

Additionally, summary statistics for the safety analysis described in Section 4.5.1 will be summarized by RVO type (BRVO and CRVO/HRVO). This includes AEs, TEAEs, SAEs, including ocular TEAEs in the study eye and non-ocular TEAEs, as well as serious ocular TEAEs in the study eye and serious non-ocular TEAEs.

#### 4.7 Interim Analyses and Data Monitoring Committee

No interim analyses in the sense of a group-sequential or adaptive design are planned.


An analysis of all data up to and including Week 36, including the primary efficacy analysis, will be performed once all participants have completed Week 36 or have discontinued the study prematurely.

A final analysis of all data, including the key-secondary analysis, will be conducted after all participants have completed the study at Week 64 or have discontinued prematurely.

A Data Monitoring Committee (DMC) that operates independently will convene periodically to assess the ongoing masked and unmasked safety data of study participants and make recommendations regarding continuation or termination of the study based on these evaluations. The DMC's operations are governed by a charter that outlines the frequency of meetings, procedures for monitoring safety (among other things), and reporting requirements to the sponsor. No adjustments to the alpha level will be made in regard to the DMC's analyses as there is no expectation of early stopping for overwhelming efficacy.

A Steering Committee will maintain close communication with the DMC, however, only masked data will be shared or discussed. Additional information about this can be found in the study protocol.

## 4.8 Changes to Protocol-planned Analyses

Since the population attribute in the estimand definition should be in reference to the target population, the population attribute in the primary and secondary estimand definition was revised from

Adult participants with treatment-naïve macular edema secondary to RVO

to

• Adult **patients** with treatment-naïve macular edema secondary to RVO.

It has been stated in the CSP Section 9.3.2.3 that an additional sensitivity analysis will be performed to account for important protocol deviations that may potentially affect efficacy for the main analysis of the primary endpoint as described in Section 4.2.2. However, it should be noted that additional ICEs may only be considered for the primary analysis, as stated in Section 4.1.8. Therefore, the sensitivity analysis will not be performed, as it is deemed obsolete in light of any additional ICEs considered for the primary analysis.

Furthermore, the definition of the FAS, as specified in the CSP Section 9.2, has been revised, as described in Section 3.

## 5. Sample Size Determination

The sample size calculation is based on the primary efficacy estimand and its endpoints, change from baseline in BCVA measured by the ETDRS letter score at Week 36.


The details of the sample size calculations can be found in Section 9.5 of the study protocol.

## **6.** Supporting Documentation

### 6.1 Appendix 1: Population characteristics

In general, variables defined in this section will have descriptive statistics presented by treatment group and overall. For continuous variables, presentation will include number of observations, mean, standard deviation, minimum, median, and maximum. For categorical variables, presentation will include number and percentage of subjects. Listings will be provided as appropriate.

### 6.1.1 Demographics and baseline characteristics

All demographic and baseline characteristics will be summarized by treatment group and overall. The descriptive statistics will be presented for the FAS and SAF.

Demographic and baseline assessments to be summarized will include:

- Age at enrollment
- Categorized age:  $< 55 \text{ years}, \ge 55 \text{ to} < 65 \text{ years}, \ge 65 \text{ years to} < 75 \text{ years}, \ge 75 \text{ years}$
- Sex: male, female
- Geographic region: Japan vs. APAC vs Europe vs America
- Ethnicity: Not Hispanic or Latino, Hispanic or Latino
- Race (only subgroups with sufficient sample size)
- Weight (kg)
- Height (cm)
- Body mass index (BMI in kg/m²)
- BMI ( $\leq$  25 kg/m², 25 kg/m² < BMI  $\leq$  30 kg/m², 30 kg/m² < BMI  $\leq$  35 kg/m², BMI > 35 kg/m²)
- Systolic blood pressure
- Diastolic blood pressure
- Baseline BCVA (ETDRS letters score)
- Baseline BCVA: < 60 letters,  $\ge 60$  letters
- Medical history of hypertension: No, Yes
- Medical history of cerebrovascular disease: No, Yes
- Medical history of ischaemic heart disease: No, Yes
- Medical history of renal impairment: Normal, Mild, Moderate, Severe
- Medical history of hepatic impairment: No, Yes
- Baseline intraocular pressure (IOP in mmHg)
- Baseline CST (in μm)


- Baseline National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25, total score)
- Baseline presence of perifoveal and parafoveal ischemia by FA
- Baseline total area of macular ischemia by FA
- Baseline presence of retinal areas of non-perfusion outside the macula by FA

#### **6.1.2 Medical History**

The medical history will be coded according to the version of Medical Dictionary for Regulatory Activities (MedDRA) available at database lock. An evaluation of medical history will be conducted through a frequency table, which will show the number of participants with medical history findings by primary system organ class (SOC) and preferred term (PT). The ocular medical or surgical history of the study eye, ocular medical or surgical history of the fellow eye, and non-ocular medical or surgical history will be summarized, respectively. All summaries will be presented for the SAF. Furthermore, a listing that includes medical history records will be provided.

## **6.1.3** Exposure and Compliance to Study Intervention

Compliance and exposure to the study intervention will be analyzed for SAF using descriptive statistics. Specifically, data up to Week 36 will be utilized for the analysis at Week 36, and data up to Week 64 will be used for the analysis at Week 64.

### 6.1.3.1 Compliance

The compliance with the study intervention will be assessed at different time points, including the first 36 weeks, and 64 weeks, or until premature discontinuation. The calculation of compliance per participant will be as follows:

Compliance = (Number of actual study interventions received during the specified period) / (Number of planned study interventions during the specified period) x = 100%.

For example, if a participant discontinues the study after Week 20 but before or at Week 24, the denominator will be 6, representing the number of planned injections until before Week 24. In the calculation of compliance, all injections, regardless of being sham or active and whether they were scheduled or unscheduled study interventions, will be considered.

The compliance data will be summarized for all periods, and a listing will be prepared to provide an overview of the compliance levels.

#### **6.1.3.2 Exposure**

For each participant, the following variables will be used to summarize the exposure to the study intervention in the study eye, including both scheduled and unscheduled interventions:

Based on actual injections:

- Total number of active injections
- Total number of sham injections
- Total amount of active study treatment (mg)


• Duration of study intervention calculated in weeks as: [(date of last study intervention prior to Week 36/ Week 64) – (date of first study intervention) +28]/7; 28 days are added because of the minimum 4-week dosing interval in the study

Based on assigned intervals as determined through IVRS based on the DRM criteria:

- Proportion of participants with specific treatment intervals (analyses up to Week 36 will only be performed for the Week 36 analysis, while analyses up to Week 64 will only be performed for the Week 64 analysis.)
  - For the 2mg group, the proportion of participants with 8 week or longer treatment interval from W32 through Week 64 (i.e., all participants extended to 8 week interval at the W32 visit for whom it was not planned to have their interval shortened to 4 week interval [according to DRM criteria] prior to Week 64).
  - o For the 8mg/3 and 8mg/5 groups, the proportion of participants with 8 week or longer treatment interval through Week 36 and Week 64 (i.e. all participants on 8 week interval for whom it was not planned to have their interval shortened to 4 week interval [according to DRM criteria] prior to Week 36 and prior to Week 64, respectively).
  - O Proportion of participants with 8 week or longer treatment interval as the last intended treatment interval at Week 36 and Week 64 in 8mg/3 and 8mg/5 groups, respectively (based on DRM criteria assessed at the last visit with active injection before Week 36 and Week 64, respectively).
  - O Proportion of participants with 8 week or longer treatment interval as the last intended treatment interval at Week 36 and Week 64 in the 2mg group, (based on DRM criteria assessed at the Week 32 visit and the last visit with active injection before Week 64, respectively).
- Proportion of participants shortening treatment intervals.
- Proportion of participants extending treatment intervals (only for Week 64 analysis).
- Proportion of participants with q4, q8, q12, or q16, as the last intended treatment interval (only for Week 64 analysis)
- Proportion of participants with q4, q8, q12, or q16, as the last completed treatment interval (only for Week 64 analysis)
- Proportion of participants shortening treatment interval at W16, W24, W32 (only for 8/3 arm)
- Proportion of participants shortening treatment interval at W24, W32 (only for 8/5 arm)
- Proportion of participants never extending treatment interval (only for Week 64 analysis)

It's important to note that these exposure variables do not consider temporary interruptions in the study intervention.

Exposure to the study intervention will be summarized for the following periods:


- From Baseline to Week 36 (excluding intervention data at Week 36) summary to be included for the Week 36 analysis
- From Baseline to Week 36 (excluding intervention data at Week 36, only participants considered as completers for Week 36) - summary to be included for the Week 36 analysis
- From Baseline to Week 64 (only participants considered as completers for Week 64) summary to be displayed for the Week 64 analysis
- From Baseline to end of the study (Week 64) summary to be displayed for the Week 64 analysis
- From Week 36 to the end of the study (Week 64) summary to be displayed for the Week 64 analysis

For each participant who received concomitant fellow eye treatment (as defined in Section 4.1.6), the following variables will be shown for SAF only:

- Total number of injections in fellow eye
- Participants without concomitant fellow eye treatment
- Participants with concomitant fellow eye treatment
  - o Aflibercept (trade name: Eylea)
  - o Bevacizumab (trade name: Avastin)
  - o Brolucizumab (trade name: Beovu)
  - o Ranibizumab (trade name: Lucentis)
  - o Faricimab (trade name: Vabysmo)
  - o Conbercept (trade name: Lumitin)
  - o Pegaptanib sodium (trade name: Macugen)

Listings will provide information on the participants' exposure duration, the number of sham and active injections, and participants who met DRM criteria will be listed separately.

#### **6.1.4** Disposition of Study Participants

The disposition of participants will be descriptively summarized in the following categories:

- The total number of participants who signed informed consent, were randomized, treated, completed study intervention and completed study for the respective analysis (Week 36 and Week 64). The summary will include all participants who gave informed consent. Participants who prematurely discontinued the study/study intervention will be summarized by reason for discontinuation.
- A summary table will include the total number and percentage of participants who qualified as FAS, SAF, and PKS (as defined in Section 3), including the reasons for exclusion from the respective analysis set.
- The disposition of participants who signed the informed consent will be summarized overall and by study site, including the date of first consent, date of last visit, and the number of participants with informed consent and in each analysis set.


- The disposition of participants and the number of sites in regions and countries will be presented for all randomized patients. Totals of all regions and within a country will be added.
- The number of participants with important protocol deviations will be presented by country and study site for all participants with signed informed consent. The number of screen failures will also be included. A second summary will show the number and percentage of participants in each protocol deviation category for the FAS. The important protocol deviations will be listed for the FAS.
- The distribution of observed ICE for the primary and key secondary estimands will be summarized by treatment group.

#### 6.1.5 Prior and Concomitant Medication

Prior and concomitant medication or therapy will be coded to Anatomical Therapeutic Chemical (ATC) classification codes according to the version of World Health Organization Drug Dictionary (WHO Drug Dictionary) available at database lock. The number and percentage of participants who took at least one prior and (new) concomitant medication and by ATC class (level 1) and subclass (level 2) will be presented for the SAF. Prior medication refers to medication taken before the start of the study drug intake, regardless of when it ended, while concomitant medication refers to medication taken during the treatment phase, between the first and last study drug intake, regardless of when it started or ended. Prior and concomitant medication for all medications will be summarized. A listing including reason for use, start and end dates and dosage information will be provided for the SAF. Participants with prior and concomitant medication will be summarized for all medications. The treatment of the fellow eye (as defined in Section 4.1.6) will be collected as concomitant medication. A listing of all prior and concomitant medication will be provided. The definitions of concomitant medications and prior medications will be used as defined above.


## 6.2 Appendix 2: Pre-defined Laboratory Abnormalities

Table 6-1: Pre-defined laboratory abnormalities

| Payments: Pre-defined laboratory abnormalities | |
|---|---|
| Parameter | Pre-defined laboratory abnormalities for phase 2/3 studies |
| Clinical chemistry | Studios |
| ALT | > 3 ULN |
| AST | > 3 ULN |
| Alkaline Phosphatase | > 1.5 ULN |
| Total Bilirubin | > 1.5 ULN |
| Conjugated bilirubin | > 35% total bilirubin (when total bilirubin >1.5 ULN) |
| ALT and Total Bilirubin | ALT > 3 ULN and Total Bilirubin > 2 ULN |
| CPK | > 3 ULN |
| Creatinine | >= 150 umol/L (1.7 mg/dL) (Adults) |
| | ≥ 30% from baseline |
| Uric Acid | Hyperuricemia: > 408 umol/L (6.86 mg/dL) |
| | Hypouricemia: < 120 umol/L (2.02 mg/dL) |
| Blood Urea Nitrogen | > 1.5 ULN |
| Chloride | < 80 mmol/L |
| Codium | > 115 mmol/L |
| Sodium | ≤ 129 mmol/L<br>≥ 160 mmol/L |
| Potassium | < 3 mmol/L |
| Fotassium | ≥ 5.5 mmol/L |
| Total Cholesterol | >= 7.74 mmol/L (299.3 mg/dL) |
| Total Offolosteror | 7 - 7.74 mmo//E (200.0 mg/dE) |
| Triglycerides | >= 4.6 mmol/L (407.3 mg/dL) |
| Glucose | , |
| - Hypoglycaemia | Hypoglycaemia: <= 3.9 mmol/L (70.3 mg/dL) and < LLN |
| - Hyperglycaemia | >= 11.1 mmol/L (200 mg/dL, unfasted), >= 7 mmol/L (126.1 mg/dL, |
| | fasted) |
| Albumin | <= 2.5 g/dL |
| , 110 GTT1111 | 2.0 g/42 |
| Hematology | |
| WBC | < 3.0 GIGA/L (non-Black), < 2.0 GIGA/L (Black), ≥ 16.0 GIGA/L |
| Lymphocytes | > 4.0 GIGA/L |
| Neutrophils | < 1.5 GIGA/L (non-Black) |
| | < 1.0 GIGA/L (Black) |
| Monocytes | > 0.7 GIGA/L |
| Basophils | > 0.1 GIGA/L |
| Eosinophils | > 0.5 GIGA/L or > ULN if ULN ≥ 0.5 GIGA /L |
| Hemoglobin | Males: <= 11.5 g/dL (7.14 mmol/L), Females: <= 9.5 g/dL (5.9 |
| | mmol/L) Decrease from baseline >= 2.0 g/dL (1.24 mmol/L) |
| | Males: >= 18.5 g/dL (11.48 mmol/L), Females: >= 16.5 g/dL (10.24 |
| | mmol/L) |
| | , |
| Hematocrit | Males: <= 37 %, Females: <= 32 % |
| | Males: >= 55 %, Females: >= 50 % |
| RBC | ≥ 6 TERA/L |
| Platelets | < 100 GIGA/L |

LLN: lower limit of normal, ULN: upper limit of normal


### 6.3 Appendix 3: Definition of safety subgroups

In the following the definitions for subgroups based on medical history and adverse events are given.

### 6.3.1 Hypertension

Hypertension will be selected based on the PTs as described in Table 6-2 below, following the PBMQ 1275. All PTs given are based on MedDRA version 26.0 and might be subject to change in future MedDRA version.

Table 6-2: PTs for selection of "Hypertension"

#### Preferred term (MedDRA version 26.0)

Accelerated hypertension

Blood pressure ambulatory increased

Blood pressure diastolic increased

Blood pressure inadequately controlled

Blood pressure increased

Blood pressure systolic increased

Diastolic hypertension

Endocrine hypertension

Essential hypertension

Hypertension

Hypertension neonatal

Hypertensive angiopathy

Hypertensive cardiomegaly

Hypertensive cardiomyopathy

Hypertensive cerebrovascular disease

Hypertensive crisis

Hypertensive emergency

Hypertensive encephalopathy

Hypertensive end-organ damage

Hypertensive heart disease

Hypertensive nephropathy

Hypertensive urgency

Labile hypertension

Malignant hypertension

Malignant hypertensive heart disease

Malignant renal hypertension

Maternal hypertension affecting foetus

Mean arterial pressure increased

Neurogenic hypertension

Nocturnal hypertension

Orthostatic hypertension

Page kidney

Prehypertension

Renal hypertension

Renovascular hypertension

Retinopathy hypertensive

Supine hypertension

Systolic hypertension

White coat hypertension


#### 6.3.2 Intraocular inflammation

Intraocular inflammation will be defined as either PBMQ 1854 Infectious Intraocular Inflammations (Eylea) or PBMQ 1855 Non-Infectious Intraocular Inflammation (Eylea), as described in Table 6-3 below. All PTs given are based on MedDRA version 26.0 and might be subject to change in future MedDRA version.

Table 6-3: PTs for selection of "Intraocular Inflammation"

### Preferred term (MedDRA version 26.0)

Anterior chamber fibrin

Anterior chamber cell

Anterior chamber flare

Anterior chamber inflammation

Aqueous fibrin

Autoimmune uveitis

Candida endophthalmitis

Chorioretinitis

Choroiditis

Cyclitis

Endophthalmitis

Eye infection bacterial

Eye infection chlamydial

Eye infection fungal

Eye infection intraocular

Eye infection staphylococcal

Eye infection

Eye inflammation

Hypopyon

Infectious iridocyclitis

Infective iritis

Infective uveitis

Iridocyclitis

Iritis

Mycotic endophthalmitis

Necrotising retinitis

Non-infectious endophthalmitis

Noninfective chorioretinitis

Pseudoendophthalmitis

Uveitis

Vitreal cells

Vitreous fibrin

Vitritis

#### 6.3.3 Nasal mucosal events

Nasal mucosal events will be defined as PBMQ - SMQ\_90001902 Nasal Mucosal Events (Eylea), as described in Table 6-4 below. All PTs given are based on MedDRA version 26.0 and might be subject to change in future MedDRA version.


Table 6-4: PTs for selection of "Nasal mucosal events"

#### Preferred term (MedDRA version 26.0)

Epistaxis
Nasal inflammation
Nasal mucosal erosion
Nasal mucosal ulcer
Nasal ulcer

## 6.3.4 Medical history of cerebrovascular disease (e.g. CVA / Stroke)

Defined by MSSO SMQ 20000060 'Central nervous system vascular disorders as described in Table 6-5 below. All PTs given are based on MedDRA version 26.0 and might be subject to change in future MedDRA version.

Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease"

#### Preferred Term (MedDRA version 26.0)

Agnosia

Amaurosis fugax

Amyloid related imaging abnormalities

Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits

Amyloid related imaging abnormality-oedema/effusion

Angiogram cerebral abnormal

Aphasia

Balint's syndrome

Basal ganglia haematoma

Basal ganglia haemorrhage

Basal ganglia infarction

Basal ganglia stroke

Basilar artery aneurysm

Basilar artery occlusion

Basilar artery perforation

Basilar artery stenosis

Basilar artery thrombosis

Benedikt's syndrome

Blood brain barrier defect

Brachiocephalic arteriosclerosis

Brachiocephalic artery occlusion

Brachiocephalic artery stenosis

Brain hypoxia

Brain injury

Brain stem embolism

Brain stem haematoma

Brain stem haemorrhage

Brain stem infarction


Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease"

#### Preferred Term (MedDRA version 26.0)

Brain stem ischaemia

Brain stem microhaemorrhage

Brain stem stroke

Brain stem thrombosis

Brain stent insertion

**CADASIL** 

CARASIL syndrome

CSF bilirubin positive

CSF red blood cell count positive

Capsular warning syndrome

Carotid aneurysm rupture

Carotid angioplasty

Carotid arterial embolus

Carotid arteriosclerosis

Carotid artery aneurysm

Carotid artery bypass

Carotid artery disease

Carotid artery dissection

Carotid artery dolichoectasia

Carotid artery insufficiency

Carotid artery occlusion

Carotid artery perforation

Carotid artery restenosis

Carotid artery stenosis

Carotid artery stent insertion

Carotid artery stent removal

Carotid artery thrombosis

Carotid endarterectomy

Carotid revascularisation

Central nervous system haemorrhage

Central nervous system vasculitis

Central pain syndrome

Cerebellar artery occlusion

Cerebellar artery thrombosis

Cerebellar atherosclerosis

Cerebellar embolism

Cerebellar haematoma

Cerebellar haemorrhage

Cerebellar infarction

Cerebellar ischaemia

Cerebellar microhaemorrhage


Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease"

#### Preferred Term (MedDRA version 26.0)

Cerebellar stroke

Cerebral amyloid angiopathy

Cerebral aneurysm perforation

Cerebral aneurysm ruptured syphilitic

Cerebral arteriosclerosis

Cerebral arteriovenous malformation haemorrhagic

Cerebral arteritis

Cerebral artery embolism

Cerebral artery occlusion

Cerebral artery perforation

Cerebral artery restenosis

Cerebral artery stenosis

Cerebral artery stent insertion

Cerebral artery thrombosis

Cerebral capillary telangiectasia

Cerebral cavernous malformation

Cerebral circulatory failure

Cerebral congestion

Cerebral cyst haemorrhage

Cerebral endovascular aneurysm repair

Cerebral gas embolism

Cerebral haematoma

Cerebral haemorrhage

Cerebral haemorrhage foetal

Cerebral haemorrhage neonatal

Cerebral haemosiderin deposition

Cerebral hypoperfusion

Cerebral infarction

Cerebral infarction foetal

Cerebral ischaemia

Cerebral microangiopathy

Cerebral microembolism

Cerebral microhaemorrhage

Cerebral microinfarction

Cerebral reperfusion injury

Cerebral revascularisation

Cerebral septic infarct

Cerebral small vessel ischaemic disease

Cerebral thrombosis

Cerebral vascular occlusion

Cerebral vasoconstriction


## Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease"

#### Preferred Term (MedDRA version 26.0)

Cerebral venous sinus thrombosis

Cerebral venous thrombosis

Cerebral ventricular rupture

Cerebrovascular accident

Cerebrovascular accident prophylaxis

Cerebrovascular arteriovenous malformation

Cerebrovascular disorder

Cerebrovascular insufficiency

Cerebrovascular pseudoaneurysm

Cerebrovascular stenosis

Charcot-Bouchard microaneurysms

Chronic cerebrospinal venous insufficiency

Claude's syndrome

Congenital cerebrovascular anomaly

Congenital hemiparesis

Delayed ischaemic neurological deficit

Diplegia

Dural arteriovenous fistula

Dysarthria

Embolic cerebellar infarction

Embolic cerebral infarction

Embolic stroke

Epidural haemorrhage

Extra-axial haemorrhage

Extradural haematoma

Extradural haematoma evacuation

Extraischaemic cerebral haematoma

Foetal cerebrovascular disorder

Foville syndrome

Haemorrhage intracranial

Haemorrhagic cerebellar infarction

Haemorrhagic cerebral infarction

Haemorrhagic stroke

Haemorrhagic transformation stroke

Heidelberg classification

Hemianaesthesia

Hemiasomatognosia

Hemiataxia

Hemidysaesthesia

Hemihyperaesthesia

Hemihypoaesthesia


Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease"

#### Preferred Term (MedDRA version 26.0)

Hemiparaesthesia

Hemiparesis

Hemiplegia

Hunt and Hess scale

Hypertensive cerebrovascular disease

Hypoxic-ischaemic encephalopathy

Inner ear infarction

Internal capsule infarction

Internal carotid artery deformity

Intra-cerebral aneurysm operation

Intracerebral haematoma evacuation

Intracranial aneurysm

Intracranial artery dissection

Intracranial haematoma

Intracranial haemorrhage neonatal

Intracranial tumour haemorrhage

Intraventricular haemorrhage

Intraventricular haemorrhage neonatal

Ischaemic cerebral infarction

Ischaemic stroke

Lacunar infarction

Lacunar stroke

Lateral medullary syndrome

Lateropulsion

Malignant middle cerebral artery syndrome

Medullary compression syndrome

Meningorrhagia

Metabolic stroke

Migrainous infarction

Millard-Gubler syndrome

Modified Rankin score decreased

Modified Rankin score increased

Monoparesis

Monoplegia

Moyamoya disease

NIH stroke scale abnormal

NIH stroke scale score decreased

NIH stroke scale score increased

**Paralysis** 

**Paraparesis** 

Paraplegia


Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease"

#### Preferred Term (MedDRA version 26.0)

Paresis

Perinatal stroke

Periventricular haemorrhage neonatal

Pituitary apoplexy

Pituitary haemorrhage

Post cardiac arrest syndrome

Post procedural stroke

Post stroke depression

Posthaemorrhagic hydrocephalus

Precerebral arteriosclerosis

Precerebral artery aneurysm

Precerebral artery dissection

Precerebral artery embolism

Precerebral artery occlusion

Precerebral artery thrombosis

Primary familial brain calcification

Pseudo-occlusion of internal carotid artery

Putamen haemorrhage

Quadriparesis

Quadriplegia

Reversible cerebral vasoconstriction syndrome

Reversible ischaemic neurological deficit

Right hemisphere deficit syndrome

Ruptured cerebral aneurysm

Septic cerebral embolism

Sigmoid sinus thrombosis

Sneddon's syndrome

Spinal artery embolism

Spinal artery thrombosis

Spinal cord haematoma

Spinal cord haemorrhage

Spinal cord infarction

Spinal cord ischaemia

Spinal epidural haematoma

Spinal epidural haemorrhage

Spinal stroke

Spinal subarachnoid haemorrhage

Spinal subdural haematoma

Spinal subdural haemorrhage

Spinal vascular disorder

Spinal vessel congenital anomaly


Table 6-5: PTs for selection of medical history of "Cerebrovascular Disease"

#### Preferred Term (MedDRA version 26.0)

Stroke in evolution

Subarachnoid haematoma

Subarachnoid haemorrhage

Subarachnoid haemorrhage neonatal

Subclavian steal syndrome

Subdural haematoma

Subdural haematoma evacuation

Subdural haemorrhage

Subdural haemorrhage neonatal

Superficial siderosis of central nervous system

Superior sagittal sinus thrombosis

Susac's syndrome

Thalamic infarction

Thalamus haemorrhage

Thrombotic cerebral infarction

Thrombotic stroke

Transient ischaemic attack

Transverse sinus thrombosis

Vascular encephalopathy

Vascular stent occlusion

Vascular stent stenosis

Vein of Galen aneurysmal malformation

Vertebral artery aneurysm

Vertebral artery arteriosclerosis

Vertebral artery dissection

Vertebral artery occlusion

Vertebral artery perforation

Vertebral artery stenosis

Vertebral artery thrombosis

Vertebrobasilar dolichoectasia

Vertebrobasilar insufficiency

Vertebrobasilar stroke

Visual agnosia

Visual midline shift syndrome

Weber's syndrome

#### 6.3.5 Medical history of ischaemic heart disease (e.g., myocardial infarction)

PBMQ SMQ\_90001278 'Medical history of myocardial infarction (VEGF Trap-Eye)' is defined by selected PTs only (from MSSO SMQs below):

• 20000043: Ischaemic heart disease (MSSO SMQ)


#### • 20000047: Myocardial infarction (MSSO SMQ)

as described in Table 6-6 below. All PTs given are based on MedDRA version 26.0 and might be subject to change in future MedDRA version.

Table 6-6: PTs for selection of medical history of "Ischaemic Heart Disease"

Acute coronary syndrome

Acute myocardial infarction

Angina pectoris

Angina unstable

Anginal equivalent

Arterial revascularisation

Arteriogram coronary abnormal

Arteriosclerosis coronary artery

Arteriospasm coronary

Cardiac perfusion defect

Cardiac ventricular scarring

Chronic coronary syndrome

Computerised tomogram coronary artery abnormal

Coronary angioplasty

Coronary arterial stent insertion

Coronary artery bypass

Coronary artery compression

Coronary artery disease

Coronary artery dissection

Coronary artery embolism

Coronary artery insufficiency

Coronary artery occlusion

Coronary artery reocclusion

Coronary artery restenosis

Coronary artery stenosis

Coronary artery surgery

Coronary artery thrombosis

Coronary brachytherapy

Coronary bypass stenosis

Coronary bypass thrombosis

Coronary endarterectomy

Coronary no-reflow phenomenon

Coronary ostial stenosis

Coronary revascularisation

Coronary steal syndrome

Coronary vascular graft occlusion

Coronary vascular graft stenosis

ECG electrically inactive area


Table 6-6: PTs for selection of medical history of "Ischaemic Heart Disease"

#### Preferred Term (MedDRA version 26.0)

ECG signs of myocardial infarction

ECG signs of myocardial ischaemia

Electrocardiogram PR segment depression

Electrocardiogram PR segment elevation

Electrocardiogram ST segment abnormal

Electrocardiogram ST segment depression

Electrocardiogram ST segment elevation

Electrocardiogram ST-T segment abnormal

Electrocardiogram ST-T segment depression

Electrocardiogram ST-T segment elevation

External counterpulsation

Haemorrhage coronary artery

Infarction

Ischaemic cardiomyopathy

Ischaemic contracture of the left ventricle

Kounis syndrome

Myocardial hypoperfusion

Myocardial hypoxia

Myocardial infarction

Myocardial ischaemia

Myocardial necrosis

Myocardial reperfusion injury

Myocardial stunning

Papillary muscle infarction

Percutaneous coronary intervention

Periprocedural myocardial infarction

Positive vessel remodelling

Post angioplasty restenosis

Post procedural myocardial infarction

Postinfarction angina

Prinzmetal angina

Scan myocardial perfusion abnormal

Silent myocardial infarction

Stent patency maintenance

Stress cardiomyopathy

Subclavian coronary steal syndrome

Subendocardial ischaemia

Vascular device occlusion

Vascular graft occlusion

Vascular graft restenosis

Vascular graft stenosis

Table 6-6: PTs for selection of medical history of "Ischaemic Heart Disease"

#### Preferred Term (MedDRA version 26.0)

Vascular graft thrombosis

Vascular stent occlusion

Vascular stent stenosis

Ventricular compliance decreased

Wellens' syndrome

# 6.3.6 Medical history of renal impairment

Renal impairment is defined by creatinine clearance (CrCl) values.

Categories for renal impairment:

- CLCR >80ml/min (normal),
- CLCR >50-80ml/min (mild),
- CLCR >30-50 ml/min (moderate),
- CLCR <=30ml/min or 'requiring dialysis' (severe).

CLCR will be calculated using baseline values (creatinine, age, weight, sex) using the Cockcroft-Gault equation:

Males: CLCR = (140-age)\*body weight / (72\*creatinine)

Females: CLCR = (140-age)\*body weight\*0.85 / (72\*creatinine)

PBMQ SMQ\_90001274 'Medical History of renal impairment requiring dialysis (VEGF Trap-Eye)' is defined by PT from Table 6-7. All PTs given are based on MedDRA version 26.0 and might be subject to change in future MedDRA version.

Table 6-7: PTs for selection of medical history of renal impairment requiring dialysis

#### Preferred Term (MedDRA version 26.0)

Continuous haemodiafiltration

Dialysis

Dialysis device insertion

Haemodialysis

Haemofiltration

Peritoneal dialysis

Removal of renal transplant

Renal replacement therapy

Renal transplant


# 6.3.7 Medical history of hepatic impairment

Defined by MSSO SMQ: Hepatic disorders 20000005 excluding sub-SMQ 20000018: Pregnancy-related hepatic disorders as described in Table 6-8 below. All PTs given are based on MedDRA version 26.0 and might be subject to change in future MedDRA version.

Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

5'nucleotidase increased

AST to platelet ratio index increased

AST/ALT ratio abnormal

Accessory liver lobe

Acquired antithrombin III deficiency

Acquired factor IX deficiency

Acquired factor V deficiency

Acquired factor VIII deficiency

Acquired factor XI deficiency

Acquired hepatocerebral degeneration

Acquired protein S deficiency

Acute graft versus host disease in liver

Acute hepatic failure

Acute hepatitis B

Acute hepatitis C

Acute on chronic liver failure

Acute yellow liver atrophy

Adenoviral hepatitis

Alagille syndrome

Alanine aminotransferase abnormal

Alanine aminotransferase increased

Alcoholic encephalopathy

Alcoholic liver disease

Allergic hepatitis

Alloimmune hepatitis

Ammonia abnormal

Ammonia increased

Anorectal varices

Anorectal varices haemorrhage

Anti factor X activity abnormal

Anti factor X activity decreased

Anti factor X activity increased

Anti-liver cytosol antibody type 1 positive

Antithrombin III decreased

**Ascites** 

Aspartate aminotransferase abnormal

Aspartate aminotransferase increased


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

**Asterixis** 

Asymptomatic viral hepatitis

Autoimmune hepatitis

**Bacterascites** 

Benign hepatic neoplasm

Benign hepatobiliary neoplasm

Benign recurrent intrahepatic cholestasis

Bile output abnormal

Bile output decreased

Biliary ascites

Biliary cirrhosis

Biliary fibrosis

Bilirubin conjugated abnormal

Bilirubin conjugated increased

Bilirubin excretion disorder

Bilirubin urine present

Biopsy liver abnormal

Blood alkaline phosphatase abnormal

Blood alkaline phosphatase increased

Blood bilirubin abnormal

Blood bilirubin increased

Blood bilirubin unconjugated increased

Blood cholinesterase abnormal

Blood cholinesterase decreased

Blood fibrinogen abnormal

Blood fibrinogen decreased

Blood thrombin abnormal

Blood thrombin decreased

Blood thromboplastin abnormal

Blood thromboplastin decreased

Bromosulphthalein test abnormal

Cardiohepatic syndrome

Cerebrohepatorenal syndrome

Child-Pugh-Turcotte score abnormal

Child-Pugh-Turcotte score increased

Cholaemia

Cholangiosarcoma

Cholestasis

Cholestatic liver injury

Cholestatic pruritus

Chronic graft versus host disease in liver

Chronic hepatic failure


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Chronic hepatitis

Chronic hepatitis B

Chronic hepatitis C

Cirrhosis alcoholic

Coagulation factor IX level abnormal

Coagulation factor IX level decreased

Coagulation factor V level abnormal

Coagulation factor V level decreased

Coagulation factor VII level abnormal

Coagulation factor VII level decreased

Coagulation factor X level abnormal

Coagulation factor X level decreased

Coagulation factor decreased

Coma hepatic

Complications of transplanted liver

Computerised tomogram liver abnormal

Congenital absence of bile ducts

Congenital hepatic fibrosis

Congenital hepatitis B infection

Congenital hepatitis C infection

Congenital hepatobiliary anomaly

Congenital hepatomegaly

Congenital viral hepatitis

Congestive hepatopathy

Cryptogenic cirrhosis

Cystic fibrosis hepatic disease

Cytokeratin 18 increased

Cytomegalovirus hepatitis

Deficiency of bile secretion

Diabetic hepatopathy

Dilatation intrahepatic duct congenital

Drug-induced liver injury

**Duodenal varices** 

Fatty liver alcoholic

Flood syndrome

Focal nodular hyperplasia

Foetor hepaticus

Galactose elimination capacity test abnormal

Galactose elimination capacity test decreased

Gallbladder varices

Gamma-glutamyltransferase abnormal

Gamma-glutamyltransferase increased


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Gastric variceal injection

Gastric variceal ligation

Gastric varices

Gastric varices haemorrhage

Gastrooesophageal variceal haemorrhage prophylaxis

Gianotti-Crosti syndrome

Glutamate dehydrogenase increased

Glycocholic acid increased

Glycogen storage disease type I

Glycogen storage disease type III

Glycogen storage disease type IV

Glycogen storage disease type VI

Graft versus host disease in liver

Granulomatous liver disease

Guanase increased

HBV-DNA polymerase increased

Haemangioma of liver

Haemorrhagic ascites

Haemorrhagic hepatic cyst

Hepaplastin abnormal

Hepaplastin decreased

Hepatectomy

Hepatic adenoma

Hepatic amoebiasis

Hepatic angiosarcoma

Hepatic artery flow decreased

Hepatic atrophy

Hepatic calcification

Hepatic cancer

Hepatic cancer metastatic

Hepatic cancer recurrent

Hepatic cancer stage I

Hepatic cancer stage II

Hepatic cancer stage III

Hepatic cancer stage IV

Hepatic candidiasis

Hepatic cirrhosis

Hepatic cyst

Hepatic cyst infection

Hepatic cyst ruptured

Hepatic cytolysis

Hepatic echinococciasis


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Hepatic encephalopathy

Hepatic encephalopathy prophylaxis

Hepatic enzyme abnormal

Hepatic enzyme decreased

Hepatic enzyme increased

Hepatic failure

Hepatic fibrosis

Hepatic fibrosis marker abnormal

Hepatic fibrosis marker increased

Hepatic function abnormal

Hepatic gas gangrene

Hepatic haemangioma rupture

Hepatic hamartoma

Hepatic hydrothorax

Hepatic hypertrophy

Hepatic hypoperfusion

Hepatic infection

Hepatic infection bacterial

Hepatic infection fungal

Hepatic infection helminthic

Hepatic infiltration eosinophilic

Hepatic lesion

Hepatic lipoma

Hepatic lymphocytic infiltration

Hepatic mass

Hepatic necrosis

Hepatic neoplasm

Hepatic neuroendocrine tumour

Hepatic pain

Hepatic perfusion disorder

Hepatic sarcoma

Hepatic sequestration

Hepatic steato-fibrosis

Hepatic steatosis

Hepatic vascular resistance increased

Hepatic venous pressure gradient abnormal

Hepatic venous pressure gradient increased

Hepatitis

Hepatitis A

Hepatitis A antibody abnormal

Hepatitis A antibody positive

Hepatitis A antigen positive


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Hepatitis A immunity confirmed

Hepatitis A virus test positive

Hepatitis B

Hepatitis B DNA assay positive

Hepatitis B DNA increased

Hepatitis B antibody abnormal

Hepatitis B antibody positive

Hepatitis B antigen positive

Hepatitis B core antibody positive

Hepatitis B core antigen positive

Hepatitis B e antibody positive

Hepatitis B e antigen positive

Hepatitis B immunity confirmed

Hepatitis B reactivation

Hepatitis B surface antibody positive

Hepatitis B surface antigen positive

Hepatitis B virus test positive

Hepatitis C

Hepatitis C RNA increased

Hepatitis C RNA positive

Hepatitis C antibody positive

Hepatitis C core antibody positive

Hepatitis C virus test positive

Hepatitis D

Hepatitis D RNA positive

Hepatitis D antibody positive

Hepatitis D antigen positive

Hepatitis D virus test positive

Hepatitis E

Hepatitis E RNA positive

Hepatitis E antibody abnormal

Hepatitis E antibody positive

Hepatitis E antigen positive

Hepatitis E immunity confirmed

Hepatitis E virus test positive

Hepatitis F

Hepatitis G

Hepatitis H

Hepatitis acute

Hepatitis alcoholic

Hepatitis cholestatic

Hepatitis chronic active


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Hepatitis chronic persistent

Hepatitis fulminant

Hepatitis infectious mononucleosis

Hepatitis mumps

Hepatitis neonatal

Hepatitis non-A non-B

Hepatitis non-A non-B non-C

Hepatitis post transfusion

Hepatitis syphilitic

Hepatitis toxic

Hepatitis toxoplasmal

Hepatitis viral

Hepatitis viral test positive

Hepato-lenticular degeneration

Hepatobiliary cancer

Hepatobiliary cancer in situ

Hepatobiliary cyst

Hepatobiliary disease

Hepatobiliary infection

Hepatobiliary neoplasm

Hepatobiliary scan abnormal

Hepatoblastoma

Hepatoblastoma recurrent

Hepatocellular carcinoma

Hepatocellular damage neonatal

Hepatocellular foamy cell syndrome

Hepatocellular injury

Hepatomegaly

Hepatopulmonary syndrome

Hepatorenal failure

Hepatorenal syndrome

Hepatosplenic abscess

Hepatosplenic candidiasis

Hepatosplenomegaly

Hepatosplenomegaly neonatal

Hepatotoxicity

Hereditary haemochromatosis

Herpes simplex hepatitis

Hyperammonaemia

Hyperbilirubinaemia

Hyperbilirubinaemia neonatal

Hypercholia


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Hyperfibrinolysis

Hypertransaminasaemia

Hypoalbuminaemia

Hypocoagulable state

Hypofibrinogenaemia

Hypoprothrombinaemia

Hypothrombinaemia

Hypothromboplastinaemia

Icterus index increased

Immune-mediated cholangitis

Immune-mediated hepatic disorder

Immune-mediated hepatitis

Increased liver stiffness

International normalised ratio abnormal

International normalised ratio increased

Intestinal varices

Intestinal varices haemorrhage

Intrahepatic portal hepatic venous fistula

Ischaemic hepatitis

Jaundice

Jaundice cholestatic

Jaundice hepatocellular

Jaundice neonatal

Kayser-Fleischer ring

Kernicterus

Leucine aminopeptidase increased

Liver abscess

Liver and pancreas transplant rejection

Liver carcinoma ruptured

Liver dialysis

Liver disorder

Liver function test abnormal

Liver function test decreased

Liver function test increased

Liver induration

Liver injury

Liver iron concentration abnormal

Liver iron concentration increased

Liver opacity

Liver operation

Liver palpable

Liver sarcoidosis


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Liver scan abnormal

Liver tenderness

Liver transplant

Liver transplant failure

Liver transplant rejection

Liver-kidney microsomal antibody positive

Lupoid hepatic cirrhosis

Lupus hepatitis

Magnetic resonance imaging hepatobiliary abnormal

Magnetic resonance proton density fat fraction measurement

Mitochondrial aspartate aminotransferase increased

Mixed hepatocellular cholangiocarcinoma

Mixed liver injury

Model for end stage liver disease score abnormal

Model for end stage liver disease score increased

Molar ratio of total branched-chain amino acid to tyrosine

Multivisceral transplantation

Necrolytic acral erythema

Neonatal cholestasis

Neonatal hepatomegaly

Nodular regenerative hyperplasia

Non-alcoholic fatty liver

Non-alcoholic steatohepatitis

Non-cirrhotic portal hypertension

Ocular icterus

Oedema due to hepatic disease

Oesophageal varices haemorrhage

Omental oedema

Osteopontin increased

Parenteral nutrition associated liver disease

Perihepatic discomfort

Perinatal HBV infection

Peripancreatic varices

Periportal oedema

Peritoneal fluid protein abnormal

Peritoneal fluid protein decreased

Peritoneal fluid protein increased

Peritoneovenous shunt

Pneumobilia

Polycystic liver disease

Porphyria acute

Porphyria non-acute


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Portal fibrosis

Portal hypertension

Portal hypertensive colopathy

Portal hypertensive enteropathy

Portal hypertensive gastropathy

Portal pyaemia

Portal shunt

Portal shunt procedure

Portal tract inflammation

Portal vein cavernous transformation

Portal vein dilatation

Portal vein flow decreased

Portal vein pressure increased

Portal venous system anomaly

Portopulmonary hypertension

Primary biliary cholangitis

Progressive familial intrahepatic cholestasis

Protein C decreased

Protein S abnormal

Protein S decreased

Prothrombin level abnormal

Prothrombin level decreased

Prothrombin time abnormal

Prothrombin time prolonged

Prothrombin time ratio abnormal

Prothrombin time ratio increased

Radiation hepatitis

Regenerative siderotic hepatic nodule

Renal and liver transplant

Retinol binding protein decreased

Retrograde portal vein flow

Reye's syndrome

Reynold's syndrome

Schistosomiasis liver

Small-for-size liver syndrome

Spider naevus

Splenic artery embolisation

Splenic varices

Splenic varices haemorrhage

Splenorenal shunt

Splenorenal shunt procedure

Spontaneous bacterial peritonitis


Table 6-8: PTs for selection of medical history of "Hepatic Impairment"

#### Preferred term (MedDRA version 26.0)

Spontaneous intrahepatic portosystemic venous shunt

Steatohepatitis

Stomal varices

Subacute hepatic failure

Sugiura procedure

Sustained viral response

Thrombin time abnormal

Thrombin time prolonged

Total bile acids increased

Transaminases abnormal

Transaminases increased

Ultrasound liver abnormal

Urine bilirubin increased

Urobilinogen urine decreased

Urobilinogen urine increased

Varices oesophageal

Varicose veins of abdominal wall

Viral hepatitis carrier

Weil's disease

White nipple sign

Withdrawal hepatitis

X-ray hepatobiliary abnormal

Yellow skin

Zieve syndrome

## 6.4 Appendix 4: Handling of Questionnaires

## 6.4.1 NEI-VFQ-25 Sub-scale Scores and Total Score

The calculation for NEI-VFQ-25 sub-scale scores and total score will be performed according to The National Eye Institute (2000). The algorithm is then: As a preparation of the VFQ-25 calculation, the items of the questionnaire will be recoded according to Table 6-9. In the further calculations, only the recoded item values will be used. For the recoded values, they generally represent the best possible result as "100" and the worst possible result as "0".


Table 6-9: Recoding of NEI-VFQ 25 items

| Item no. | Original response to | Recoded item |
|---|---|---|
| 1, 3, 4, 15c <sup>(a)</sup> | 1 | 100 |
| | 2 | 75 |
| | 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| 2 | 1 | 100 |
| | 2 | 80 |
| | 3 | 60 |
| | 4 | 40 |
| | 5 | 20 |
| | 6 | 0 |
| 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 16a | 1 | 100 |
| -, - | 2 | 75 |
| | 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| | 6 | * |
| 17, 18, 19, 20, 21, 22, 23, 24, 25 | 1 | 0 |
| ,,,,,,,, | 2 | 25 |
| | 3 | 50 |
| | 4 | 75 |
| | 5 | 100 |

<sup>(</sup>a) Item 15c has four-response levels but is expanded to a five-levels using item 15b: if 15b="1", then 15c="0" / if 15b=("2" or "3"), then 15c="missing"

For the VFQ questionnaire, 12 sub-scales will be evaluated (see Table 6-10), and 11 of these sub-scales will be included in the total VFQ score.

Table 6-10: Sub-scales of the NEI-VFQ 25 score

| Sub-scale no. | Sub-scale | | Number of items | (Recoded)<br>items to be<br>averaged | Sub-scale<br>included in total<br>scale |
|---|---|---|---|---|---|
| 1 | General Health | 1 | | 1 | No |
| 2 | General Vision | 1 | | 2 | Yes |
| 3 | Ocular Pain | 2 | | 4, 19 | Yes |
| 4 | Near Activities | 3 | | 5, 6, 7 | Yes |
| 5 | Distance Activities | 3 | | 8, 9, 14 | Yes |
| | Vision specific: | | | | _ |
| 6 | Social Functioning | <u>j2</u> | | 11, 13 | Yes |
| 7 | Mental Health | 4 | | 3, 21, 22, 25 | Yes |
| 8 | Role Difficulties | 2 | | 17, 18 | Yes |
| 9 | Dependency | 3 | | 20, 23, 24 | Yes |
| 10 | Driving | 3 | | 15c, 16, 16a | Yes |
| 11 | Color vision | 1 | | 12 | Yes |
| 12 | Peripheral Vision | 1 | | 10 | Yes |

<sup>\*</sup> Here, Response choice "6" indicates that the person does not perform the activity because of non-vision-related problems. If this choice is selected, the item is coded as "missing".


For a single sub-scale, the value will be determined as the average of the non-missing recoded item values assigned to this sub-scale. A sub-scale value will only be assessed as missing if all items for this sub-scale have "missing" as a result.

The total score is calculated as the arithmetic mean of all non-missing sub-scales (except General Health):

$$total\ result = \frac{(sum\ of\ non\ - missing\ sub\ -\ scale\ values)}{Total\ number\ of\ sub\ -\ scales\ with\ non\ -\ missing\ result}$$

Due to this calculation approach, the total result will be non-missing if at least one sub-scale result is non-missing.

# 6.5 Appendix 5: Strategies for displaying Summary Statistics

The strategies for displaying summary statistics based on the primary estimand and for utilizing imputation of missing data with LOCF are presented in Table 6-11 and Table 6-12, respectively.

Table 6-11: Strategies for displaying Summary Statistics in line with the primary estimand

| Intercurrent event | Analysis |
|---|---|
| | and discontinuation of study: non-observed data beyond discontinuation of study intervention will not be included in the summary statistics |
| | and continuation of study: observed data beyond last active injection (that was administered before the premature discontinuation of study intervention) + current treatment interval +5 days will be excluded from summary statistics |
| Use of a prohibited medication (as per section 4.1.7) before Week 36 | Observed data beyond first administration of the prohibited medication in study eye will be excluded from the summary statistics |
| Missed active injection resulting in an actual injection interval up to 4 weeks longer than planned | All observed data will be <u>included</u> in the summary statistics |
| Missed active injection resulting in an actual injection interval more than 4 weeks longer that planned | Observed data beyond last active injection (that was nadministered before the first missed active injection) + current treatment interval +5 days will be excluded from the summary statistics |


Table 6-12: Strategies for displaying Summary Statistic using imputation of missing values with LOCF.

| Intercurrent event | Analysis |
|---|---|
| Premature discontinuation of study intervention for any reason before Week 36 | and discontinuation of study: non-observed data beyond discontinuation of study intervention will be imputed using LOCF |
| | and continuation of study: observed data beyond last active injection (that was administered before the premature discontinuation of study intervention) + current treatment interval +5 days will be excluded from summary statistics and imputed by LOCF |
| Use of a prohibited medication (as per section 4.1.7) before Week 36 | Observed data beyond first administration of the prohibited medication in study eye will be excluded from the summary statistics and resulting missing data will be imputed by LOCF. |
| Missed active injection resulting in an actual injection interval up to 4 weeks longer than planned | All observed data will be <u>included</u> in the summary statistics |
| Missed active injection resulting in an actual injection interval more than 4 weeks longer that planned | Observed data beyond last active injection (that was nadministered before the first missed active injection) + current treatment interval +5 days will be excluded from summary statistics and imputed by LOCF |

# 6.6 Appendix 6: Identification of intake of prohibited medications and cases of prohibited procedures

To identify any intake of prohibited medications (see Section 4.1.7), Table 6-13 provides a list of corresponding WHO drug names and record numbers. The list is based on the specific medications mentioned in Section 4.1.7 and additionally on observed concomitant medications during study conduct meeting the definition in Section 4.1.7 as of finalization of this statistical analysis plan. The list may be updated before unmasking and this would be documented in a separate document.

Table 6-13: Preliminary list of prohibited medication by drug names (may be updated before unmasking of the data)

| WHO Drug Name | WHO Drug<br>Record Number | WHO Drug Sequence<br>Number 1 | WHO Drug Sequence<br>Number 2 |
|---|---|---|---|
| Aflibercept | 062254 | 01 | any |
| Bevacizumab | 015552 | 01 | any |
| Brolucizumab | 088687 | 01 | any |
| Conbercept | 073395 | 01 | any |


| Faricimab | 156766 | 01 | any |
|-------------------------|--------|----|-----|
| Pegaptanib sodium | 022285 | 02 | any |
| Ranibizumab | 020889 | 01 | any |
| Ocriplasmin | 079085 | 01 | 001 |
| Dexamethasone (Ozurdex) | 000160 | 01 | 404 |

As for prohibited procedures (also see Section 4.1.7), cases of vitrectomy surgery will be identified from the Surgical, Diagnostic and Therapeutic Procedure(s) page using the standardized procedure name "Vitrectomy". Cases of retinal laser photocoagulation for the treatment of RVO will be identified based on a dedicated protocol deviation (PD) category (PD Term: Subject received laser therapy for treatment of their macular edema secondary to RVO in the study eye.).

## 7. References

- 1. Gasparyan SB, Folkvaljon F, Bengtsson O, Buenconsejo J, Koch GG. Adjusted win ratio with stratification: Calculation methods and interpretation. *Statistical Methods in Medical Research*. 2021;30(2):580-611. doi:10.1177/0962280220942558
- 2. Efron, B., and Tibshirani, R. J. (1993). An Introduction to the Bootstrap. New York, NY: Chapman and Hall. doi: 10.1007/978-1-4899-4541-9
- 3. Heitjan, F., and Little, R. J. A. (1991). "Multiple Imputation for the Fatal Accident Reporting System." Journal of the Royal Statistical Society, Series C 40:13–29
- 4. Holz FG, Roider J, Ogura Y, Korobelnik JF, Simader C, Groetzbach G, et al. VEGF Trap-Eye for macular oedema secondary to central retinal vein occlusion: 6-month results of the phase III GALILEO study. Br J Ophthalmol. 2013;97(3):278-84.
- 5. Ratitch B, Lipkovich I, O'Kelly M. Combining Analysis Results from Multiply Imputed Categorical Data. PharmaSUG 2013 Paper SP0.
- 6. Rogers S, McIntosh RL, Cheung N, Lim L, Wang JJ, Mitchell P, et al. The prevalence of retinal vein occlusion: pooled data from population studies from the United States, Europe, Asia, and Australia. Ophthalmology. 2010;117(2):313-9.e1.
- 7. Rubin D E. Multiple Imputation for Nonresponse in Surveys. Wiley. 1987
- 8. Schenker, N., and Taylor, J. M. G. (1996). "Partially Parametric Techniques for Multiple Imputation." Computational Statistics and Data Analysis 22:425–446.
- 9. Stokes ME, Davis CS, Koch GG. Categorical Data Analysis Using SAS, Third Edition. SAS Institute, 2012